# Ketamine Tolerated Dose to Prevent Postpartum Depression and Pain after Cesarean Delivery (PREPARE 1)

Protocol Number: STUDY22100018 Version Date: 05/29/2024 7.0 Version Number: IND Sponsor: University of Pittsburgh Principal Investigator: Grace Lim, MD, MSc IND Number: IND 142105 NCT Number: NCT05907213 Source of Funding: National Institute of Mental Health: R01MH134538

# History of Protocol Versions:

| Version | Date | Sections Changed | Rationale for the Change |
|---|---|---|---|
| 1.0 | April 26, 2023 | N/A | N/A |
| 2.0 | May 30, 2023 | 5.2 inclusion criteria 5.4 payment plan 6.4 storage in lockbox 7.4 patient safety | IRB comment response |
| 3.0 | June 6, 2023 | 5.4 payment plan | |
| 4.0 | September 12, 2023 | Various | Update consistency with MOP DSMB edits |
| 5.0 | September 22, 2023 | 1<br>5.2 | Study population clarification Updated inclusion wording |
| 6.0 | | Protocol Overview Section 4 | Updated wording for clarity Revised wording to make timing of assessments clearer |
| | | Section 5.2 | Revised inclusion criteria to clarify only cesarean delivery, removal of neuraxial morphine restriction as it is not germane to the primary study objectives, specified term delivery definition |
| | December 7, 2023 | Section 5.3 | Revised exclusion criteria to clarify patient undergoing general anesthesia to match wording in other documents; other wording modification to match wording in institutional protocol; removed contraindication to NSAID as it is not germane to primary study objective |

| | | Section 7.1 | Updated screening procedures to reflect workflow optimization |
|---|---|---|---|
| | | Section 7.6 | Corrected a spelling error |
| | | Section 8.2 | Deleted "risks of withholding<br>breastfeeding for 60 hours" as we<br>are not asking women to<br>withhold breastfeeding |
| | | Section 9.2 | Spelling error |
| 7.0 | | Appendix 3 | Corrected to include protocollisted assessments at postpartum week 12, which is Day 84, Visit 13 |
| | | Appendix 2 | Corrected RASS and vital signs to line up with protocol text LSD >8 cutoff for PI notification and bedside check to enhance safety and facilitate direct event attributions |
| | May 16, 2024 | Figure 1 | Corrected to line up with protocol text for RASS, side effect assessments and postpartum assessments |
| | | Section 3.4.1, 6.3, Table 1 of Section 6.2 | DLT event definition revised to include complete infusion cessation due to intolerable side effect acceptability ratings by patient. Table now specifies events that qualify as DLT in accordance with revised DLT definition |

| Section 6.2 | Added grace period range +15<br>minutes for maintenance infusion<br>dose adjustment times |
|---|---|
| Sections 3.4.1, 6.3, 9.1, 12.3, Table 1 of Section 6.2 | Reduced systolic blood pressure cutoff from 190mmHg to 160mmHg in accordance with DSMB recommendations and to be more aligned with systolic blood pressure cutoffs in the pregnant and postpartum population |
| Section 6.6 | Clarified rescue medication protocol for nausea/vomiting |

# Contents

| 1 | Pr | otocol Overview | 1 |
|---|-----------------|---------------------------------------|-----|
| | 1.1 | Study Schema | . 2 |
| 2 | Ba | ckground and Rationale | 3 |
| | 2.1 | Background | . 3 |
| | 2.2 | Rationale | . 4 |
| 3 | - | potheses, Objectives and Endpoints | |
| | 3.1 | Hypotheses | |
| | 3.2 | 5 51 | |
| | 3.3 | Objectives | |
| | 3.3 | .1 Primary Objective: | . 4 |
| | 3.3 | .2 Secondary Objective | . 4 |
| | 3.3 | .3 Exploratory Objectives | . 5 |
| | 3.4 | Endpoints | . 5 |
| | 3.4 | .1 Primary Endpoint | . 5 |
| | 3.4 | .2 Secondary Endpoints | . 5 |
| 4 | | search Design | |
| 5 | | ıman Subjects | |
| | 5.1 | Subject Population | |
| | 5.2 | Inclusion Criteria | |
| | 5.3 | Exclusion Criteria | |
| | 5.4 | Recruitment Methods | |
| | 5.5 | Screen Failures | |
| 6 | <b>St</b> : 6.1 | Udy Drug | |
| | 6.2 | Study Drug Preparation and Dispensing | |
| | 6.3 | Dose Delays and Modifications | |
| | 6.4 | Study Drug Storage and Accountability | |
| | 6.5 | Prohibited Medications | |
| | 6.6 | Rescue Medications | 15 |
| 7 | | search Activities | |
| | 7.1 | Screening Procedures | 19 |

| | 7.2 | Study Entry Procedures | . 19 |
|---|---|---|---|
| | 7.3 | Study Drug Administration | . 19 |
| | 7.4 | Safety Assessments/Procedures During Treatment | . 20 |
| | 7.5 | Safety Assessments/Procedures During Follow-up | . 20 |
| | 7.6 | End of Study Safety and Efficacy Assessments/Procedures | . 20 |
| 8 | Po | tential Risks and Benefits | 20 |
| | 8.1 | Reasonably Foreseeable Risks Related to Study Drug | . 21 |
| | 8.2 | Reasonably Foreseeable Risks Related to Research Interventions | . 21 |
| | 8.3 | Potential Benefits | . 22 |
| 9 | Pr | otection Against Risks | 22 |
| | 9.1 | Management of drug related toxicity | . 22 |
| | 9.2 | Management of research related risks | . 22 |
| 1( | ) Ad | lverse Events and Serious Adverse Events | 23 |
| | 10.1 | Severity | . 24 |
| | 10.2 | Relatedness | . 25 |
| | 10.3 | Expectedness | . 25 |
| | 10.4 | Reporting Serious Adverse Events | . 26 |
| 1: | L W | ithdrawal of Subjects and Stopping Rules | 26 |
| | 11.1 | Adverse Events Requiring Discontinuation | . 26 |
| | 11.2 | Other Criteria Requiring Discontinuation | . 27 |
| | 11.3 | Clinical Trial Stopping Rules | . 28 |
| 12 | 2 Sta | atistical Analysis | 28 |
| | 12.1 | General Approach | . 28 |
| | 12.2 | Sample Size Determination | . 29 |
| | 12.3 | Analysis of Primary Endpoint | . 29 |
| | 12.4 | Analysis of Secondary Endpoints | . 29 |
| 13 | 3 Da | ıta and Safety Monitoring | 29 |
| | 13.1 | Data Safety Monitoring Plan | |
| | 13.2 | Parameters to be Monitored | . 30 |
| | 13.3 | Frequency of Monitoring | . 31 |
| | 13.4 | Clinical Monitoring | . 31 |
| | 13.5 | Data and Safety Monitoring Board | 31 |

| 14 Regulatory, Ethical, and Study Oversight | 32 |
|---|---|
| 14.1 IRB Approval | |
| 14.2 Informed Consent Procedures | 32 |
| 14.3 Protocol Deviations | 33 |
| 15 References | 35 |
| Appendix 1 – Surveys Measures | 48 |
| Appendix 2 – Schedule of Perinatal, Surgical, and Infusion-Specific Research Activities | |
| Appendix 3 – Schedule of Postpartum Research Activities | |

# **ABBREVIATIONS AND ACRONYMS**

| AE | Adverse Event |
|--------|------------------------------------------------------|
| ADL | Activities of Daily Living |
| ASA PS | American Society of Anesthesiologist Physical Status |
| AUC | Area Under Curve |
| CD | Cesarean Delivery |
| CFR | Code of Federal Regulations |
| Cmax | Peak concentration of "drug" |
| CRF | Case Report Form |
| Css | Concentration of "drug" at Steady State |
| DHHS | Department of Health and Human Services |
| DLT | Dose Limiting Toxicity |
| DSMB | Data Safety Monitoring Board |
| EPDS | Edinburgh Postnatal Depression Scale |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HIPAA | Health Insurance Portability and Accountability Act |
| IB | Investigator's Brochure |
| ICH | International Conference on Harmonization |
| IDE | Investigational Device Exemption |
| IDS | Investigational Drug Service |
| IND | Investigational New Drug Application |
| IRB | Institutional Review Board |
| ITT | Intention-To-Treat |
| IV | Intravenous |
| MDD | Major Depressive Disorder |
| MTD | Maximum Tolerate Dose |
| NCT | National Clinical Trial |
| NIH | National Institutes of Health |
| NMDA | N-Methyl-D-Aspartate Receptor |
| PCP | Phencyclidine |
| PD | Pharmacodynamics |
| PI | Principal Investigator |
| PK | Pharmacokinetic |
| PPD | Postpartum Depression |
| PSS | Perceived Stress Scale |
| RASS | Richmond Agitation Sedation Scale |
| REDCap | HIPAA compliant data management software |
| RID | Relative Infant Dose |
| SAE | Serious Adverse Event |
| SSRI | Selective Serotonin Reuptake Inhibitor |
| UPMC | University of Pittsburgh Medical Center |

# 1 Protocol Overview

| Study Description | The purpose of this study is to identify a tolerable dose for postpartum ketamine infusion using a maximum tolerated dose (MTD) 3+3 design. A loading dose over 1 hour will be the MTD variable to be tested, as our data suggest that ketamine side effects occur with the loading dose. |
|---|---|
| Study Population: | Patients having cesarean delivery (CD) who are either: 1) planning not to breastfeed; or 2) are receiving ketamine as part of clinical care, will be enrolled. Ketamine will be started in postpartum patients, after cord clamping. |
| Planned Sample Size: | The projected sample size will be a maximum of 12 patients with complete primary outcome data within the MTD 3+3 design. |
| Participating Institutions (if a multicenter clinical trial) | N/A |

# 1.1 Study Schema

Figure 1. Assessment timeline for MTD study and follow-up assessments



Figure 2. MTD dosing schematic for PREPARE 1.



# 2 Background and Rationale

# 2.1 Background

A lack of data on new pain treatments in pregnancy and lactation puts 1.2 million US women having cesarean delivery (CD) every year at risk for poor pain control, depressed mood, and poor recovery<sup>7,8</sup>. Despite high individual variability in pain after CD<sup>6,9</sup>, current CD treatments ignore the multidimensionality of pain, including the influence of mood on pain. NMDA receptor antagonists like ketamine significantly reduce postoperative pain and opioid use by up to 40%<sup>10</sup>. In addition to its analgesic effects, a single dose of IV ketamine has been shown to rapidly reduce depressive symptoms by 50% and remission rates 43-77%<sup>86</sup> in non-obstetric populations. Evidence of successful post-surgical pain management and rapid reduction of depressive symptoms render ketamine a great candidate for post-CD pain management and potential reduction of PPD symptomology.

Ketamine at sub-anesthetic doses is effective in post-surgical acute pain management, with long-lasting analgesia. Many trials (non-obstetric) have shown ketamine effectiveness for post-operative analgesia $^{94.96}$ . Available postpartum ketamine studies have focused on various doses (ranging 0.1-0.5 mg/kg, single doses, infusions) for efficacy $^{16-18,66}$ , but have not emphasized side effects. Although high doses of ketamine induce psychomimetic effects, low doses, such as in the current proposal, can reduce pain without side effects $^{10,78}$  and potentially reduce pain intensity for 1 year after a single dose (effect size 0.61, 95% CI 0.40 – 0.80) $^{97}$ .

In addition to its analgesic effects, ketamine use for depression treatment promotes fast, effective depression symptom reductions, a robust effect occurs from 4-72 hours post-infusion (0.5 mg/kg over 40 min) in patients with MDD; this dose is commonly used for depression<sup>87</sup>. The antidepressant effect lasts beyond psychotomimetic symptoms, which peak during the infusion and return to baseline within 1-2 hours<sup>86</sup>. These findings contrast traditional antidepressants whereby only 1/3 of patients become symptom-free after 7 weeks of treatment with SSRI.<sup>85</sup> A widely cited trial of 205 ketamine doses (0.5mg/kg, 40 min) for depression concluded ketamine was, "safe and well- tolerated" but did not probe patient acceptability of side effects<sup>33</sup>. Dose-dependent side effects are common, with a high incidence of vertigo, nausea, sedation, and dissociation in intranasal dosing to plasma levels similar to an IV dose of 0.5 mg/kg over 40min<sup>88</sup>. These dose-dependent side effects preclude widespread use in the peripartum population. Identifying ketamine dose tolerability in a post-CD population has the potential to improve treatment of postoperative pain as well as mood-related outcomes of chronic pain such as comorbid onset of PPD. This work will

Defining postpartum ketamine PK is critical to understanding the potential role of ketamine for PPD prevention, and to understanding the plasma ketamine concentration time profile with its maximum tolerated dose. There are no PK/PD models for ketamine-induced side effects or analgesia, although there are isolated reports of ketamine side effects with plasma concentrations. Available trials that conclude ketamine is "well tolerated" did not query patient perspectives in acceptability<sup>33</sup>. The duration of ketamine exposure may be important as well, given that subcutaneous administration may have greater antidepressant duration than intravenous administration of the same dose, despite lower

peak plasma concentrations in subcutaneous administration<sup>19</sup>. These knowledge gaps are significant because they limit patient-centered acceptability of ketamine and a finer understanding of its potential effective utility for PPD prevention. Because ketamine is metabolized by CYP3A and CYP2B6 (increased activity in pregnancy and immediately after delivery)<sup>34</sup>, and because pregnancy induces sensitivity to anesthetics, it is critical in this project to identify a tolerable dose of postpartum ketamine and the perioperative factors impacting its PK.

#### 2.2 Rationale

Defining postpartum ketamine tolerable doses and ketamine PK is critical to understanding the potential role of ketamine for PPD prevention, and to understanding the plasma ketamine concentration time profile with its maximum tolerated dose. There are no PK/PD models for ketamine-induced side effects or analgesia, although there are isolated reports of ketamine side effects with plasma concentrations. Available trials that conclude ketamine is "well tolerated" did not query patient perspectives in side effect acceptability<sup>33</sup>. The duration of ketamine exposure may be important as well, given that subcutaneous administration may have greater antidepressant duration than intravenous administration of the same dose, despite lower peak plasma concentrations in subcutaneous administration<sup>19</sup>. These knowledge gaps are significant because they limit patient-centered acceptability of ketamine and a finer understanding of its potential effective utility for PPD prevention. Because ketamine is metabolized by CYP3A and CYP2B6 (increased activity in pregnancy and immediately after delivery)<sup>34</sup>, and because pregnancy induces sensitivity to anesthetics, it is critical in this project to identify a tolerable dose of postpartum ketamine and the perioperative factors impacting its PK.

# 3 Hypotheses, Objectives and Endpoints

# 3.1 Hypotheses

# 3.2 Primary Hypothesis

The purpose of this study is to identify a tolerable dose for postpartum ketamine infusion using a maximum tolerated dose (MTD) 3+3 design. A loading dose over 1 hour will be the MTD variable to be tested, as our data suggest that ketamine side effects occur with the loading dose.

Our working hypothesis, based on our preliminary PK and safety data and that of Loo et al [19], is that a 12-hr IV ketamine infusion of 0.05 mg/kg/hour is the MTD.

# 3.3 Objectives

#### 3.3.1 Primary Objective:

Quantify maximum tolerable dose of postpartum ketamine infusion post-cesarean delivery.

# 3.3.2 Secondary Objective

Quantify *side effect* acceptability of low-dose ketamine infusion in peripartum people.

### 3.3.3 Exploratory Objectives

Measure maternal pain and depression in this cohort before and after cesarean delivery until 12weeks postpartum.

# 3.4 Endpoints

# 3.4.1 Primary Endpoint

Maximum Tolerated Dose (MTD). The MTD will be defined as the dose at which fewer than 33% of patients experience a DLT defined by intolerability.

Tolerability (dichotomous Yes/No)

Tolerability (YES) will be defined as: lack of adverse events (adverse event defined as: severe unresolved hemodynamic effect: systolic blood pressure <80 or >160, heart rate <40 or >120).

Lack of Tolerability will be defined as presence of any adverse event (i.e., severe unresolved hemodynamic effect: systolic blood pressure <80 or >160, heart rate <40 or >120).<sup>33</sup>

A **DLT** event is defined by complete infusion cessation due to intolerable side effect acceptability ratings by patient, OR the experience of an intolerable event as defined above. The escalation of dosing will be as noted in Figure 2 and is based on a modified Fibonacci sequence  $^{101,102}$  with smaller proportional increases in dose in the escalation scheme. Escalations occur until 2 in a cohort of 3 to 6 experiences DLT (i.e., until  $\geq$ 33% of patients experience DLT at that dose). The dose **below** this level estimates the MTD.

Participants will be classified as having had a DLT if any of the following conditions are met:

- Persisting (i.e., unresolved after 3 consecutive measurements within a 15-minute interval)
  hemodynamic side effects defined as below and despite treatments or minimizing
  infusion rates as specified.
  - Systolic blood pressure <80 or >160
  - Heart rate <40 or >120
- Complete infusion cessation due to intolerable side effect acceptability ratings by patient

Primary Outcomes will be measured at a minimum of every 4-hours from the start of the ketamine infusion (t = 0) for 24-hours (12-hours post infusion cessation). Additional assessments will be administered between the 4-hour measurements if any adverse event or side effect is noted by the patient.

# 3.4.2 Secondary Endpoints

Patient-reported *side effect* acceptability ratings, defined below Peripartum pain scores, defined in Appendix 1

Peripartum depression scores, defined by Edinburgh Postnatal Depression Score (EPDS)

# Side Effect Acceptability Ratings

Any reported side effects are rated by patients. Patient reported side effects (i.e., dizziness, lightheadedness, bad dreams, nausea, vomiting, itchiness, and hallucinations: all dichotomous outcomes) will be evaluated based on patient-specific reports of how "acceptable" or "unacceptable" the side effects are for continued or future use of the study medication. Patient-reported acceptability is defined based on theoretical framework of acceptability<sup>103</sup> and focused on constructs of Burden ("Would experiencing side effects keep you from participating in this intervention (ketamine) again?" yes/no) and Affective Attitude ("Based on your experience with this medication, would you be willing to participate in this intervention (ketamine) again?" yes/no).

- 1. Acceptability is the absence of patient-centered unacceptable side effects. Patients with side effects who report that the side effects were "acceptable" on digital diary will be counted as having confirmed **side effect** acceptability ratings, regardless of the presence of any side effects to the ketamine dose. Patient-reported acceptability is defined as a "yes" to Affective Attitude with a "no" to Burden.
- 2. Unacceptability is any patient report of unacceptable side effects, defined as any positive response on the digital side effect diary rated unacceptable by the patient. Either a negative response to Attitude, or a positive response to Burden, will define patient unacceptability.

# 4 Research Design

This is an open-label maximum tolerated dose (MTD) 3+3 design. 101,102

# Protocol Overview.

Patients will respond to surveys prior to and following cesarean delivery regarding their current pain and mood. Patients will begin study procedures in the third trimester of pregnancy, within approximately one week of scheduled cesarean delivery, until 12-weeks postpartum.

Preoperative weight and vital signs will be measured, and baseline inventories completed (Figure 1; refer to section 1.1). After delivery, cord clamping and declaration of clinical stability by the anesthesiologist (typically~5-15 min after delivery; ±30 minutes), a loading infusion of ketamine 0.05 mg/kg/hour will begin for the first 3-patients in the study. Vital signs and side effect symptomology will be measured 15, 30, and 60 minutes (±5 minutes) after infusion start, and at 4, 8, 10, 12, 16, and 24 hours (±30 minutes) after infusion start. Plasma samples will be collected at 1, 6, 10, and 12 hours (±30 minutes) after infusion. Any report of adverse events or side effects will trigger a blood draw for analysis and correlation of these symptoms to plasma levels of ketamine within the 12-hour infusion. All assessments have been timed to coincide with timing intervals of typical post-CD clinical care interventions. Patients dosing after the first three patients will proceed based on the MTD protocol in Figure 2; refer to section 1.1.

MTD dosing protocol.

A loading dose and maintenance infusion strategy will be used (Figure 2; in section 1.1). MTD to be tested will focus on the initial loading dose used to achieve a higher plasma concentration in a brief period. Ketamine dose will not exceed sub-anesthetic ranges (≤0.2mg/kg/hr<sup>78</sup>). The maintenance rate of 0.05mg/kg/hr is based on our preliminary data suggesting tolerability, and on data suggesting that this rate might yield adequate plasma concentrations necessary for the treatment of depression. The first set of 3 patients will receive a loading infusion of ketamine 0.05 mg/kg/hr for the first data. The decision to escalate the loading infusion dose, enter 3 more at the same level, or stop, will not occur until 3 patients complete the 0.05 mg/kg/hr protocol. A **DLT** event is defined in section 3.4.1.

# 5 Human Subjects

# 5.1 Subject Population

The maximum tolerated dose (MTD) 3+3 design encompasses blocks of 3 patients allocated to dosing schematics. In this study, we have 4 dosing schematics to be tested. Therefore, a minimum number of 6 and maximum number of 12 patients will participate in this trial.

#### 5.2 Inclusion Criteria

- Cesarean delivery
- Adults 18 years and older
- Term delivery ≥ 37 weeks gestation anticipated at time of delivery
- ASA PS 2 or 3
- •
- \_
- One of the following must be met for inclusion:
  - Not planning to breastfeed
  - o Ketamine use indicated for pain management plan.

#### 5.3 Exclusion Criteria

- Patient going under general anesthesia for cesarean delivery
- Allergy to study medication (ketamine)
- ASA PS 4 +
- Contraindications to neuraxial anesthesia
- Preterm delivery (<37 weeks gestation)</li>
- Anticipated fetal-neonatal complex care plan as indicated in the patient's chart
- Patient history of ketamine or PCP abuse
- Patient history of schizophrenia or psychosis
- Patient history of liver or renal insufficiency
- Patient history of uncontrolled hypertension, chest pain, arrhythmia, head trauma, or intracranial hypertension, uncontrolled thyroid disease, or other contraindications to ketamine
- Participating in another pain intervention trial

- Pre-eclampsia with severe features
- Hemodynamic instability
- Contraindicated medications use:
  - o Oral antihypertensive medications (exclusion: hypertensive disorders of pregnancy)
  - o Intravenous magnesium (exclusion: pre-eclampsia with severe features)
  - Ketamine, phencyclidine, psilocybins, or any other psychedelics (exclusion: ketamine or PCP abuse)
  - Lithium, valproate, carbamazepine, lamotrigine, haloperidol, chlorpromazine, fluphenazine, aripiprazole, clozapine, or other typical or atypical
  - o antipsychotic medications (exclusion: schizophrenia or psychosis)

#### 5.4 Recruitment Methods

The current process for research recruitment is that the research anesthesia team will review charts for all patients presenting for cesarean delivery or who are likely to present for a cesarean delivery in the labor and delivery rooms. Prenatal records will indicate patients planning not to breastfeed. During prenatal anesthesiology evaluations, the anesthesiology team will identify patients who are including ketamine infusion as part of their pain management care. Research staff will contact patients to explain the availability of the study to the patient meeting eligibility criteria.

Additional methods of recruitment include directly approaching potential subjects (in-person), the use of Email/Listserv/Electronic Mailing List, use of Flyers/Posters or Brochures in provider offices and clinics, use of Pitt+Me university research registry portal, and patient/participant referrals.

Patients will be eligible if they are receiving ketamine as part of their clinical care, and these typically include patients with a history of complex pain, history of chronic pain with or without treatment, current everyday smokers, patients with opioid or substance use disorder, and patients who have a documented history of treated or untreated anxiety, depression, or trauma.

Eligible patients will be notified of their eligibility to participate in the study by clinical and research staff. Should the patient wish to hear more, the study coordinator will discuss study participation. Questions will be answered, and time will be afforded to patients per the Informed Consent Procedures outlined, to minimize risks of coercion or undue influence.

Upon completion of the baseline inventories and the ketamine infusion and blood collection, patients will receive a payment of \$750 (see Appendix 4 for payment details). Upon completion of the postpartum weekly surveys, payments of up to \$150 will be made at both 6- and 12-weeks postpartum.

*In-Hospital Encounter*Baseline inventories

| Complete infusion and all blood draws | \$ 750.00 |
|--------------------------------------------|----------------|
| Postpartum Encounters | |
| Complete all weekly surveys @ \$25.00/week | |
| Complete weekly surveys for 6 weeks | up to \$150.00 |
| Complete weekly surveys for weeks 7-12 | up to \$150.00 |
| <b>Grand Total</b> | \$ 1,050.00 |

#### 5.5 Screen Failures

Participants who are consented to participate in the third trimester of pregnancy, may be withdrawn from the study protocol before, during, or following the cesarean surgery if events arise such as to preclude them from participating in the remainder of the study. These participants will be considered "Screening Failures". The following list is non-comprehensive, but represents the most likely scenarios:

- Vaginal or non-cesarean delivery
- Development of exclusion-based criteria prior to cesarean surgery (i.e., severe preeclampsia, preterm delivery, NICU assessment likely, etc.)
- Severe complications during labor and/or delivery whereby the PI and/or patient's surgeon recommend a change in therapeutic response.

Withdrawn participants will be replaced at a proportion of 1:1. Procedures are as follows:

- Study personnel and investigators will be notified.
- Written documentation of withdrawal and reason for withdrawal will be noted per IRB protocol.
- Study personnel, investigators, and pharmacy will be informed of the need for replacement of pharmaceuticals due to participant withdrawal.
- Subsequent data to be collected from the withdrawn participant will be restricted to the minimum amount necessary to continue to monitor safety, i.e., side effect diary including questions of sedation, LSD short form, dizziness, lightheadedness, bad dreams, nausea, vomiting, pruritus, hallucinations.

# 6 Study Drug

Ketalar (Ketamine) (C13H16ClNO, 2-(2-chlorophenyl)-2-(methylamino) cyclohexan-1-one) is a cyclohexanone derivative with known analgesic and anesthetic properties. It inhibits biogenic amine uptake, binds opioid receptors, and inhibits N-methyl D-aspartate (NMDA) receptors.

Ketamine will be used for post-cesarean delivery analgesia. Specifically, it will be evaluated for its role in pain reduction, opioid reduction, and improved pain outcomes. In the non-obstetric surgical population, modalities such as intravenous ketamine are well-recognized as effective adjuncts in opioid-reduction strategies for postoperative pain. Ketamine is used off-label as standard clinical care in perioperative pain management for patients with a history of complex pain such as people with chronic

pain (treated or untreated), a history of or current symptoms of depression and anxiety, current smokers, and women with opioid or substance use disorders.

Ketamine is an approved drug or biologic being evaluated for a new indication, population, route of administration, or dosage level not specified in the FDA approved labeling.

#### 6.1 Dose Selection

Safety and Efficacy: Preclinical studies, including studies on animals, and clinical studies, including studies on non-pregnant women, have been conducted and provide reassuring data on minimal potential risks to postpartum women. [45 CFR 46.204 (a)]. The selected reference list below demonstrates experience with this drug in dosing regimens matching or exceeding the currently proposed dosing, in both pregnant and postpartum people. The data support low risks to this population. In the dosing regimen that we describe which is "sub-anesthetic" (i.e.,  $\leq 0.2 \text{ mg/kg/hr}$ , lower than the anesthetic dosing regimens), we expect that the risks are sufficiently low to justify studying it in this fashion.

#### Selected Relevant References

- Suppa E, Valente A, Catarci S, Zanfini BA, Draisci G. A study of low-dose S-ketamine infusion as "preventive" pain treatment for cesarean section with spinal anesthesia: benefits and side effects. Minerva Anestesiol. 2012 Jul;78(7):774-81.
- Joel S, Joselyn A, Cherian VT, Nandhakumar A, Raju N, Kaliaperumal I. Low-dose ketamine infusion for labor analgesia: A double-blind, randomized, placebo controlled clinical trial. Saudi J Anaesth. 2014 Jan;8(1):6-10.
- Sen S, Ozmert G, Aydin ON, Baran N, Caliskan E. The persisting analgesic effect of low-dose intravenous ketamine after spinal anaesthesia for caesarean section. Eur J Anaesthesiol. 2005 Jul;22(7):518-23.
- Menkiti ID, Desalu I, Kushimo OT. Low-dose intravenous ketamine improves postoperative analgesia after caesarean delivery with spinal bupivacaine in African parturients. Int J Obstet Anesth. 2012 Jul;21(3):217-21.
- Bilgen S, Köner O, Türe H, Menda F, Fiçicioğlu C, Aykaç B. Effect of three different doses of ketamine prior to general anaesthesia on postoperative pain following Caesarean delivery: a prospective randomized study. Minerva Anestesiol. 2012 Apr;78(4):442-9.
- Heesen M, Böhmer J, Brinck EC, Kontinen VK, Klöhr S, Rossaint R, Straube S. Intravenous ketamine during spinal and general anaesthesia for caesarean section: systematic review and meta-analysis. Acta Anaesthesiol Scand. 2015 Apr;59(4):414-26.
- Bauchat JR, Higgins N, Wojciechowski KG, McCarthy RJ, Toledo P, Wong CA. Low-dose ketamine with multimodal postcesarean delivery analgesia: a randomized controlled trial. Int J Obstet Anesth. 2011 Jan;20(1):3-9.
- Reza FM, Zahra F, Esmaeel F, Hossein A. Preemptive analgesic effect of ketamine in patients undergoing elective cesarean section. Clin J Pain. 2010 Mar-Apr;26(3):223-6.

# 6.2 Study Drug Preparation and Dispensing

The study drug, ketamine, will be sourced by investigational (IDS) Pharmacy at UPMC Magee Women's Hospital. The infusions will be packaged and labeled for use in the clinical research study per pharmacy protocols and guidelines. Ketamine will be prepared by pharmacy with dosing instructions. There will be no blinding.

For on-site preparation and dispensing of the study drugs, the following procedures will be followed. The pharmacist of record will: maintain adequate records confirming receipt, expiration dates, or other disposition information on the investigational drug; they will record the name of the individual to whom the drug is shipped, date, quantity, and batch number. They will secure the drug in a locked storage area and monitor to ensure proper storage conditions; they will also complete regular inventory to assure accurate indication of stock on hand, as well as proper recording of stock received, dispensed, and returned. For the patients enrolled for open label pharmacokinetic studies, the pharmacist will generate a label prior to dispensing the study drug, including the date dispensed, quantity and expiration information, drug strength and dose; they will affix the label to the dispensed drug. For dispensing and drug disposition recording, they will record the date dispensed, patient initials or other identifiers, drug treatments, quantity dispensed, initials of dispenser, date and amount of patient returns documented in study records (i.e., returned drug that cannot be re-dispensed). Filing and all drug documentation will occur within study records, medical records, and logs.

Following the cesarean delivery, the initial drug administration (via IV infusion) will begin 15 minutes (± 30 minutes) after cord clamping and declaration of clinical/ hemodynamic stability by the case anesthesiologist after delivery. The maintenance dose will start 60 min (range: +15min) after the initial loading dose. The infusion will be completely stopped 12 hours after the start of infusion. The same infusion pump will follow the patient throughout the postoperative period for 12 hours until completion of the study drug. No manipulation of the infusion pump will occur by the patient. Adjustments to the rate will be at the discretion of the study team and can be physically made by study personnel qualified and trained in these procedures, or by clinical care providers under direct orders from the study team.

#### 6.3 Dose Delays and Modifications

All subjects will be monitored for adverse events throughout participation in this trial. Events requiring a dose delay or adjustment are described below.

#### Adverse Event, Dose Delays or Adjustments Procedures.

Contingency for lowest dose not tolerated. Our preliminary data suggests that only 1/8 (12.5%) of individuals received an infusion rate lower than 0.05mg/kg/hr due to side effects. However, these data are not representative of our study population, so it is conceivable that PK or PD for side effects may differ in the immediate postpartum setting, and that the lowest loading dose may not be tolerated. If loading dose of 0.05mg/kg/hr is not tolerated, we will follow the dose adjustments in Table 1 and Figure 3 below.

# Events that Trigger Dose Adjustment Procedures:

- Persisting unresolved hemodynamic side effects defined as Systolic blood pressure <80 or >160,
   Heart rate <40 or >120<sup>33</sup>
  - o Unresolved after 3 consecutive measurements within a 15-minute interval
- Persisting (i.e., unresolved within 1 hour of onset) side effects sedation, dizziness, lightheadedness, persistent itchiness, bad dreams, hallucinations, or other side effects that are reported as not acceptable to patients or clinicians, despite minimizing infusion rate.
- Table 1 includes procedures for dose adjustments.

# Patient Reported Side Effects Dose Delays or Adjustments

- Side Effect Acceptability ratings are defined in section 3.4.2. Patient reported side effects (i.e., dizziness, lightheadedness, bad dreams, nausea, vomiting, itchiness, and hallucinations: all are dichotomous outcomes). These side effects will be evaluated based on patient-specific reports of how "acceptable" or "unacceptable." Patients reporting side effects and rating them as "unacceptable" will follow the dose delay or adjustment described in the Table 1. If side effects are rated "acceptable" then no dose delays or adjustments will occur.
- Figure 3 Decision Chart for Acceptability Based dose revisions.

Table 1. Loading and Maintenance Dose Adjustment Procedures:

| Systolic blood pressure <80 or >160, Heart rate <40 or >120 Monitor for 5 minutes minutes for symptom resolution Monitor for 5 minutes for symptom resolution If event does not resolve Hold infusion for 5 box (e.g., 0.05mg/kg/hr) and continue infusion. If event does not resolve Hold infusion for 5 box (e.g., 0.05mg/kg/hr) and continue infusion. May D/C infusion and monitor subject for safety as | Event | 1st Action | 2 <sup>nd</sup> 1 | Action | 3rd / | Action | If event does not resolve |
|---|---|---|---|---|---|---|---|
| Pressure <80 or >160, Heart rate <40 or >120 Heart rate <40 or >1 | | | | | | | |
| monitor subject for safety as described in Section 7.4 and described in Section 7.4 and 7.5 Event qualifies as DLT | pressure <80 or >160, | labetalol or<br>hydralazine per<br>managing<br>anesthesiologist<br>Monitor for 5<br>minutes for<br>symptom | for 5 minutes -<br>symptom<br>recheck at 5 | (e.g.,<br>0.05mg/kg/hr<br>reduced to 0.025<br>mg/kg/hr) and<br>continue | for 5 minutes - symptom recheck at 5 minutes: May D/C infusion based on investigator discretion and monitor subject for safety as described in Section 7.4 and | (e.g.,<br>0.025mg/kg/hr<br>reduced to 0.013<br>mg/kg/hr) and<br>continue | minutes of unresolved hemodynamic effect: D/C infusion and monitor subject for safety as described in Section 7.4 and 7.5 Event qualifies |

| Event | 1st Action | <b>2</b> <sup>nd</sup> A | Action | 3rd A | Action | If event does not resolve |
|---|---|---|---|---|---|---|
| | | If event does<br><u>not</u> resolve | If the event<br>resolves | If event does<br><u>not</u> resolve | If the event<br>resolves | <u></u> 1650.776 |
| If RASS -2 or below,<br>OR Respiratory Rate<br>is < 8 | Hold infusion<br>for 10 minutes -<br>symptom<br>recheck every<br>10 min until<br>resolution | If no resolution within 1 hour: D/C infusion based on investigator discretion and monitor subject for safety as described in Section 7.4 and 7.5 | ↓ dose by 50% (e.g., 0.05mg/kg/hr reduced to 0.025 mg/kg/hr) and continue infusion. | If no resolution within 1 hour: D/C infusion based on investigator discretion and monitor subject for safety as described in Section 7.4 and 7.5 | ↓ dose by 50% (e.g., 0.025mg/kg/hr reduced to 0.013 mg/kg/hr) and continue infusion. | D/C infusion<br>and monitor<br>subject for<br>safety as<br>described in<br>Section 7.4 and<br>7.5<br>Event qualifies<br>as DLT |
| Dizziness,<br>lightheadedness, bad<br>dreams, persistent<br>itchiness,<br>hallucinations,<br>nausea, vomiting, or<br>other side effects<br>rated by patient as<br>Not Acceptable | Hold infusion<br>for 10 minutes -<br>symptom<br>recheck every<br>10 min until<br>resolution<br>Supportive care<br>medications in<br>9.1 | If no resolution within 1 hour: D/C infusion based on investigator discretion and monitor subject for safety as described in Section 7.4 and 7.5 | ↓ dose by 50% (e.g., 0.05mg/kg/hr reduced to 0.025 mg/kg/hr) and continue infusion. | If no resolution within 1 hour: D/C infusion based on investigator discretion and monitor subject for safety as described in Section 7.4 and 7.5 | ↓ dose by 50% (e.g., 0.025mg/kg/hr reduced to 0.013 mg/kg/hr) and continue infusion. | D/C infusion<br>and monitor<br>subject for<br>safety as<br>described in<br>Section 7.4 and<br>7.5<br>Event qualifies<br>as DLT |
| Nausea or Vomiting | Rescue medications as indicated in 6.6 Re-evaluate for symptom resolution 10 min after rescue medication Hold infusion for 10 minutes - symptom recheck every 10 min until resolution | If no resolution within 1 hour: D/C infusion based on investigator discretion and monitor subject for safety as described in Section 7.4 and 7.5 | dose by 50% (e.g., 0.05mg/kg/hr reduced to 0.025 mg/kg/hr) and continue infusion. | If no resolution within 1 hour: D/C infusion based on investigator discretion and monitor subject for safety as described in Section 7.4 and 7.5 | dose by 50% (e.g., 0.025mg/kg/hr reduced to 0.013 mg/kg/hr) and continue infusion. | D/C infusion<br>and monitor<br>subject for<br>safety as<br>described in<br>Section 7.4 and<br>7.5<br>Event qualifies<br>as DLT |

Figure 3. Dose adjustments based on patient-reported acceptability



#### 6.4 Study Drug Storage and Accountability

For on-site preparation and dispensing of the study drugs, the following procedures will be followed. The investigational drug (IDS) pharmacist of record will: maintain adequate records confirming receipt, expiration dates, or other disposition information on the investigational drug; they will record the name of the individual to whom the drug is shipped, date, quantity, and batch number. They will secure the drug in a locked storage area and monitor to ensure proper storage conditions; they will also complete regular inventory to assure accurate indication of stock on hand, as well as proper recording of stock received, dispensed, and returned. For the 24 patients enrolled for open label pharmacokinetic studies, the pharmacist will generate a label prior to dispensing the study drug, including the date dispensed, quantity and expiration information, drug strength and dose; they will affix the label to the dispensed drug. Pharmacist will generate a label prior to dispensing the study drug, including the date dispensed, quantity and expiration information; they will affix the label to the dispensed drug; they will record but not disclose on the label the drug strength and dose. For dispensing and drug disposition recording,

they will record the date dispensed, patient initials or other identifiers, drug treatments, quantity dispensed, initials of dispenser, date and amount of patient returns documented in study records (i.e., returned drug that cannot be re-dispensed). Filing and all drug documentation will occur within study records and IDS logs. During the infusion, the ketamine will be stored in a lockbox and all Magee standard of care procedures for the safety of controlled substances will be in place for the use of ketamine from the start of infusion through the end of the infusion in the postpartum unit.

#### 6.5 Prohibited Medications

Medications that will not be permitted prior to or during subject participation in the study are as follows:

- Oral antihypertensive medications (exclusion: hypertensive disorders of pregnancy)
- Intravenous magnesium (exclusion: pre-eclampsia with severe features)
- Ketamine, phencyclidine, psilocybins, or any other psychedelics (exclusion: ketamine or PCP abuse)
- Lithium, valproate, carbamazepine, lamotrigine, haloperidol, chlorpromazine, fluphenazine, aripiprazole, clozapine, or other typical or atypical antipsychotic medications (exclusion: schizophrenia or psychosis)

#### 6.6 Rescue Medications

Rescue antiemetics will be provided for patients reporting nausea or vomiting. The following medications will be used to treat nausea or vomiting at the time of patient reporting these symptoms:

- Ondansetron 4mg IVP p.r.n. nausea or vomiting or
- Dexamethasone 4-6mg IVP p.r.n. nausea or vomiting
- After a total of two doses of ondansetron or dexamethasone, additional rescue antiemetics will be given at the full discretion of anesthesiologist

# 7 Research Activities

Figure 1 (section 1.1) illustrates all encounters for measurements at the preoperative baseline, during the intraoperative period, ketamine infusion period, in the postpartum hospital stay (or until patient discharge), and the 1- to 12-week assessments of pain and depression. Study procedures will begin at enrollment pre-operatively, continue during the ketamine infusion, and hospital post-operative stay, continue weekly in the postpartum period, and end at 12-weeks postpartum.

Information collected at baseline includes maternal demographic information, prenatal pain and depressive symptomology, concurrent acute pain, and covariables such as demographic characteristics, and perceived stress. EPDS is completed twice, at least 1 week apart, prior to delivery. The baseline measures are repeated weekly in the postpartum period until 12-weeks postpartum.

During the ketamine infusion, blood samples will be taken at 1-, 6-, 10-, & 12-hours post-infusion start, as well as at the time of any adverse side effect report to assess ketamine/metabolite levels at the time of event.

### Baseline (Preoperative) Procedures.

- a. **Demographic Data and Medical History.** Demographic data will be collected through self-reported questions through the RedCap interface. Data from the medical record will be extracted and recorded by trained research associates to be entered into the RedCap interface. Individual surveys are transposed into RedCap for ease of patient use either on a tablet or paper when patients are in person, and via text or email-linked surveys for remote responses. Survey measure timepoints are described in the Appendix.
- b. **Surveys**. Patient-reported measures will occur by validated instruments delivered by paper, tablet (in hospital), or via Mosio text-based interface with data integration via REDCap. Texting and email will be used via patient-preferred cellular phone numbers and email addresses for 12-weekly postpartum assessments. Each weekly assessment will occur within ±3 days of the weekly postpartum date. Each set of patient-reported REDCap surveys, in total, is expected to last between 15- and 20-minutes, except for the postoperative timepoints which are expected to take less than 15-minutes to complete. Specific surveys and timeline of surveys will be as follows and as indicated in Table 1 and Figure 1.

### **Intraoperative Procedures:** Day of Surgery

Standardized Surgical, Anesthesia and Analgesia Protocols

Surgical personnel role will be recorded (e.g., titles such as private vs faculty obstetricians, resident, or physician assistant). Standardized spinal anesthesia and intraoperative medications will be as follows. Intraoperative medications include current clinical standards of prophylactic phenylephrine infusion to reduce hypotension and related intraoperative nausea/vomiting; ondansetron at the time of delivery for postpartum nausea/vomiting prophylaxis; and ketorolac 15-30 mg at the time of facial closure. Rescue analgesia and antiemetics will follow our existing clinical protocols.

*Spinal anesthesia medications*: bupivacaine 0.75% 1.6mL with fentanyl 10-15mcg and morphine 100-150mcg.

#### Co-medications:

- Per clinical routine, prophylactic phenylephrine infusion at 0.5 mcg/kg/min (37.5mL/hr at standard concentrations) will be started at the beginning of spinal anesthesia induction and discontinued at the time of delivery.
- Supplemental vasopressor boluses are delivered at the full discretion of the managing anesthesiology team.
- Ondansetron 4mg IVP for PONV prophylaxis
- Dexamethasone 4mg IVP for PONV prophylaxis unless contraindications
- Acetaminophen 1000mg either orally pre-operatively or IVPB at facial closure

# • Ketorolac 15-30mg IVP at facial closure

Rescue intraoperative antiemetic: Ondansetron 4mg IVP as a rescue dose as needed x1 dose; dexamethasone 4-6mg IVP as needed x1 dose; after this, additional rescue antiemetic can be given at the full discretion of the managing anesthesia team.

# Postpartum Analgesia Protocol

Postpartum analgesia protocols will be aligned with routine clinical practice at UPMC Magee-Womens Hospital. Specifically, ketorolac 30 mg IV q6h x24 hours (total of 4 doses) will be administered. After all doses of ketorolac have been given, ibuprofen 600mg q6h x24 hours will be delivered, not to be given within 6 hours of ketorolac. Acetaminophen 500-650mg q4h no more than 4000mg q24hr will be given with the first dose given on postoperative day 0. For severe breakthrough pain rated 7-10 on VAS, the Investigator will be called to assess the need to order oxycodone 5-10mg if necessary, as needed for severe breakthrough pain. The Investigator may also assess the need for parenteral rescue agents, namely hydromorphone.

### Discharge Analgesia Regimen

Consistent with current routine clinical practice at UPMC Magee, subjects will be discharged with a prescription for oxycodone 5-10mg q6h #12-20 p.r.n. severe pain. Adjustments to this regimen will be made on an individual basis based on prescriber and institutional practice changes that may arise.

# Surgical case reports.

Surgical elements will be collected from surgeons as well as data abstraction from the medical record (Table 3). Surgeons will complete the Surgeon Operative Survey (Table 2) described below:

# Table 2. Surgical Operative Survey

# Surgeon/Obstetrician Operative Survey

- 1. Reason for Cesarean Delivery
- 2. Type of Skin Incision
- 3. Type of Uterine Incision
- 4. Dissection type and inclusion of rectus
- 5. Uterine exteriorization
- 6. Bladder Flap
- 7. Any unanticipated surgical challenges?
- 8. Please rate difficulty of delivery
  - (0-10 numeric rating scale, 0 is no difficulty, 10 is the most difficult imaginable)
- 9. Please rate difficulty of overall surgery (0-10 numeric rating scale, 0 is no difficulty, 10 is the most difficult imaginable)
- 10. Please rate degree of adhesive disease (0-10 numeric rating scale, 0 is no adhesive disease, 10 is the most adhesive disease imaginable)
- 11. Please rate degree of difficulty of fetal extraction. (0-10 numeric rating scale, 0 is no adhesive disease, 10 is the most adhesive disease imaginable)
- 12. Were there any unanticipated surgical challenges encountered? (yes/no)
- 13. Did you make any intraoperative consultations to other surgeons? (yes/no)
- 14. What materials were used for Facial and Skin closure.

Table 3. Surgical data abstraction from the medical record

| Element | Where to find in EHR |
|---|---|
| Duration of surgery (min) | Cerner Surginet Operative Report |
| Surgical assist role (resident, physician assistant) | Cerner Surginet Operative Report |
| Surgical attending role (private vs faculty) | Cerner Surginet Operative Report |
| Infant weight (grams) | Cerner Surginet Operative Report |
| Apgar score 1 minute (integer 0-9) | Cerner Surginet Operative Report |
| Apgar score 5 minutes (integer 0-9) | Cerner Surginet Operative Report |
| Estimated blood loss (mL) | Cerner Surginet Operative Report<br>Cerner SA Anesthesia Record |
| Total intravenous fluids administered (mL) | Cerner SA Anesthesia Record |
| Total urine output (mL) | Cerner SA Anesthesia Record |
| MME Opioid use in postpartum days 1-3 | Cerner SA Anesthesia Record |

# Ketamine Infusion, Side Effect Measures, and Plasma Sampling Procedures.

Preoperative weight and vital signs will be measured, and baseline inventories completed (Figure 1). After delivery, cord clamping and declaration of clinical stability by the anesthesiologist (approximately 5-15 minutes after delivery, ± 30 minutes), a loading infusion of ketamine 0.05 mg/kg/hr will begin for the first 3-patients in the study. Vital signs and Richmond Agitation Scale (RASS), and self-reports of side effects will be measured 15, 30, and 60 minutes (±10 minutes) after infusion start, and at 4-8-10-12-16-24- hours (±30 minutes) after infusion start. Plasma samples will be collected at 1-6-, 10- and 12- hours (±30 minutes) after infusion start via an indwelling IV catheter to facilitate ease of access. Plasma samples at 1-6-, 10- and 12- hours after infusion start will be used to calculate Cmax, AUC, and Css and to correlate DLTs with these PK parameters. Any report of adverse events or side effects will trigger a blood draw for analysis and correlation of these symptoms to plasma levels of ketamine. All assessments have been timed to coincide with timing intervals of typical post-CD clinical care interventions. Patient dosing after the first three patients will proceed based on the MTD protocol in Section 1.1.

#### MTD Dose Adjustment Procedures.

Figure 2 (section 1.1) outlines the dosing approach. Dose adjustment procedures are outlined in section 6.3.

#### Side Effect Acceptability Ratings.

Our existing and previously tested **digital diary** will automate alerts for questions about side effects after infusion start at 15-, 30-, 60- minutes, and every 4 hours in the first 24 hours after infusion start (Figure 1, section 1.1). The diary has been tested and used by our group in previous work; alerts coincide with RASS assessments and similar timing of clinical assessments for routine CD nursing care and monitoring (i.e., is not more burdensome or intrusive to patients than routine clinical post-CD care). The digital diary will assess side effects

(i.e., dizziness, lightheadedness, bad dreams, nausea, vomiting, itchiness, and hallucinations: all dichotomous outcomes). Any positive response to any item will trigger the subject to rate their acceptability of side effects in the following way. Patient-reported acceptability is defined based on theoretical framework of acceptability<sup>103</sup> and focused on constructs of *Burden* ("Would experiencing side effects keep you from participating in this intervention (ketamine) again?" yes/no) and *Affective Attitude* ("Based on your experience with this medication, would you be willing to participate in this intervention (ketamine) again?" yes/no). Either a negative response to Attitude, or a positive response to Burden, will define patient unacceptability.

#### Side Effects.

Monitoring during the infusion will follow our clinical standards of perioperative ketamine monitoring. A maternal side effect digital diary will also be used. The digital diary has been previously developed and tested in our preliminary lactation volunteer study. The diary alerts questions to patients include the Richmond agitation-sedation scale (RASS)<sup>104</sup>, dysphoria (LSD short form<sup>105</sup>), and side effects. Automated alerts for abnormal responses go to clinical and research staff for immediate action. Any report of side effects will trigger a blood draw for analysis and correlation to measured plasma levels.

### Postpartum 12-week Follow-up Procedures.

Figure 1 (section 1.1) outlines weekly follow-up procedures. Participants will receive weekly surveys containing the questionnaires that are specified in Appendix 1. Surveys focus on pain and depression symptoms throughout the postpartum period.

# 7.1 Screening Procedures

Per our existing research procedures, patients will be screened from the Magee-Womens Hospital OB surgery schedule by dedicated trained research associates. Screening will be completed using the "Core Surgical PowerChart" and "Epic" Electronic Health Record (EHR) systems. All procedures will follow existing processes with clinicians for patient enrollment in research. Patients scheduled for CD are contacted prior to surgery by phone or in person to assess eligibility, explain the study protocol, and provide consent. Patients who are eligible within the prenatal clinics will be contacted prior to surgery in person, via a MyUPMC message or using videoconferencing to explain the study and obtain consent.

#### 7.2 Study Entry Procedures

Participants will be screened for eligibility prior to consent. Inclusion criteria and exclusion criteria are described in Sections 5.2 and 5.3.

# 7.3 Study Drug Administration

Following the cesarean delivery, the initial drug administration will be made after cord clamping and once anesthesiologist has declared hemodynamic stability (i.e., infusion starts approximately 5-15 minutes after delivery,  $\pm$  30 minutes). The infusion will be completely stopped at 12 hours after the start of infusion. The same infusion pump will follow the patient throughout the postoperative period for 12 hours until completion of the study drug. No manipulation of the infusion pump will occur by the

patient. Adjustments to the rate will be at the discretion of the study team and can be physically made by study personnel qualified and trained in these procedures, or by clinical care providers under direct orders from the study team.

### 7.4 Safety Assessments/Procedures During Treatment

Maternal monitoring during the infusion will follow our clinical standards perioperative ketamine monitoring and the standard Magee system safety precautions for administration of a controlled substance will be in place to protect from any misuse. A licensed and qualified anesthesia provider (resident, fellow, nurse anesthetists, or anesthesiologist) will be present during the first 30 minutes of the infusion and will have the option to treat blood pressures >180/100 mm Hg or heart rate >110 bpm. The study infusion will be discontinued if 3 consecutive measurements within a 15-minute interval remain above protocol-defined limits despite intervention (section 6.3). Maternal side effect symptomology monitoring will occur throughout the ketamine infusion. Automated alerts for maternal side effect responses go to clinical and research staff for immediate action. Any report of side effects will trigger a blood draw for analysis and correlation to measured plasma levels.

An independent DSMB will define frequency of monitoring of tolerability and DLT data. The severity of adverse events are classified in section 10.1

### 7.5 Safety Assessments/Procedures After Ketamine Infusion Stop

Maternal side effect monitoring following the infusion will continue at 4-hour intervals for 12-hours after the cessation of ketamine infusion. Monitoring will occur via clinical staff monitoring and via patient self-report indices of side effect symptomology (Figure 1; section 1.1).

After the study drug infusion is complete, safety and efficacy assessments consist of the following. Digital diaries will assess self-reported side effects according to the study schematic Figure 1; 1.1, until 12 hours after infusion discontinuation. Vital signs will be monitored during that same period.

#### 7.6 Safety Assessments/Procedures During Postpartum Surveys

Efficacy assessments, exploratory in nature, will consist of pain and depression symptom screening at regular intervals from one week postpartum until 12 weeks after delivery, according to the time intervals indicated in the study schematic Figure 1; 1.1. Positive screens for depression will be initiate an immediate response to the study team. The protocol for positive depression screens is presented in Appendix 4. All patients who screen positive for depression (EPDS total score > 14 or positive answer to question #10) will be contacted and receive consultation instructions.

After all study procedures are complete 12 weeks after delivery, there will be no further active assessments of safety and efficacy by study staff. Participants will continue to have access to their primary care physicians and emergency services.

#### 8 Potential Risks and Benefits

# 8.1 Reasonably Foreseeable Risks Related to Study Drug

Common side effects of ketamine are sedation, dizziness, lightheadedness, bad dreams, hallucinations, euphoria, dysphoria, nausea, vomiting. These risks are minimized by using doses below the doses that we typically see these side effects. Seriousness: mild to moderate.

Uncommon effects of ketamine include hypertension or hypotension, tachycardia, or bradycardia. These risks are minimized as much as possible by using doses below the doses that we typically see these effects. If these effects are noted, the drug will be stopped until the effects dissipate. Should the effects not dissipate, the PI will evaluate and determine whether the patient requires additional care. If these uncommon effects are experienced, an SAE log will be completed and the IDSMB and IRB notified. Seriousness: mild to moderate

# 8.2 Reasonably Foreseeable Risks Related to Research Interventions

Risks to confidentiality. There is a risk of breach of confidentiality with the screening procedures and the collection and storage of personal health information. To protect against this risk, all screening procedures will be done by study staff who have been completely trained in HIPAA/privacy procedures; all data collected will be identifiable only by a unique subject ID number, and no personal identifiers will be stored with the data. Linkage files identifying subjects will be stored only in physical records that are kept in locked files accessible only by study staff; electronic data will be handled and protected whereby any linkages between study ID number and patient identification will be separated, password protected, and stored behind the UPMC firewall. There are some cases in which a researcher is obligated or authorized by law to report mental health symptoms, such as serious threats to public health and safety. For example, if patients indicate that they are in imminent risk of harm (e.g., suicide or serious threats toward the wellbeing of others), the researchers will contact the appropriate authorities to protect patients or the public. Seriousness: mild

*Risks of inconvenience from surveys.* To minimize the inconvenience/time burden on participants associated with the survey questions, we will use an electronic (email) interface preferentially and will minimize the number of questions to strictly only the number necessary to address important aspects of our study questions. Seriousness: mild

*Risk of survey discomfort.* An uncommon risk includes inconvenience and potential emotional discomfort are risks associated with answering survey questions. Subjects will be asked to answer questions regarding pain and depression before, during, and after having their babies. Answering these questions may be viewed as an inconvenience. Seriousness: mild

*Risks of IV blood collection.* Common risks associated with blood collection include bruising or swelling at the collection sight, discomfort during venous blood draw, and infection. Seriousness: mild

Risk of sub-anesthetic ketamine infusion dose titration. Common risks include nausea, euphoria, dizziness, or lightheadedness. Seriousness: mild. Uncommon risks include temporary hypertensive event.

Seriousness: mild to moderate; uncommon risks include hallucinations or dysphoria. Seriousness: mild to moderate.

#### 8.3 Potential Benefits

The potential direct benefits to subject participation in this study is enhanced pain control, opioid reduction, closer follow-up for depression symptoms, and reduced depression risk. There are societal benefits in that there will be increased knowledge about the use of ketamine after birth to reduce depression, alleviate pain and decrease opioid use. Ultimately, the results of this study, if significant, will enable health care providers to improve the health of mothers.

### 9 Protection Against Risks

# 9.1 Management of drug related toxicity

The PI is a practicing, board-certified clinical anesthesiologist with extensive experience in the administration of this study drug under normal clinical circumstances. The study drug will be started during routine anesthesia care where monitoring is the strictest and closest, thereby enabling early detection of any safety events. The patients will remain monitored in an appropriate care environment throughout the duration of the 12-hour drug infusion, enabling timely detection and treatment of any serious events should they occur. Staff will also be trained to be familiar with common and uncommon side/adverse events for reporting.

Supportive care drugs that may be used in the event of drug related toxicity:

- Event: Persisting unresolved hemodynamic side effects defined as Systolic blood pressure <80 or >160, heart rate <40 or >120, unresolved after 3 consecutive measurements within a 15-minute interval
  - Supportive care medications:
  - Labetalol 10-20mg IVP or Hydralazine 10-25mg IVP p.r.n. hypertension at discretion of managing anesthesiologist.
- Event: Persisting side effects sedation, dizziness, lightheadedness, bad dreams, hallucinations, or other side effects that are reported as not acceptable to patient or clinicians, despite minimizing infusion rate
  - Supportive care medications:
  - o Midazolam 1-4mg IVP p.r.n. dysphoria, at discretion of managing anesthesiologist.

Refer to Section 6.8 for Rescue Drugs.

Refer to Section 6.3 of the protocol for instructions on dose delays and modifications.

# 9.2 Management of research related risks

All research interventions/activities will be conducted in private patient care areas. The collection of sensitive information about subjects is limited to the amount necessary to achieve the aims of the research, so that no unneeded sensitive information is collected.

All demographic and clinical information about the subject will be stored in an electronic password-guarded study database under the supervision of the Investigator for this protocol. The electronic system REDCap has features that can enable its use as certifiably compliant with the DFTA regulations at 21 CFR part 11 but due to the limited scope of this clinical research study, the electronic data recording system has not been certified as fully compliant. The data will be stripped of individual identifiers at the time of analysis and stored anonymously with a subject number. Information linking subject identifiers with the coded subject number will be stored under password proection on computers in locked areas, with access to the database manager. Access to the database will be limited to the data manager and staff under the supervision of the Investigator.

All staff involved in this study are properly credentialed and instructed in the areas of testing, confidentiality, and safety. All study team members will be properly trained on protocol requirements, trained in HIPAA/privacy procedures, and GCPs. Research procedures performed for study purposes will be performed by qualified individuals as evidenced by education, experience, and/or training. All members of the study team will have the required human subjects and confidentiality training, which includes information about maintaining data integrity and security. Confidentiality will be guarded using established procedures such as storing data in locked cabinets within locked offices or locked data rooms, coding CRFs and research specimens by study identification numbers rather than any personal identifying information to avoid revealing the identity of subjects, and aggregating data across participants. The key linking names and study identification numbers will be kept separately from the data sets with limited access by study personnel. Only study personnel will have access to the data sets on protected servers.

The Investigator will retain the data for the entire period of this study and will retain the specified records and reports for up to seven years after the study's publication. The Investigator may continue to use and disclose subjects' de-identified information for the purpose of this study for a minimum of seven years after final reporting or publication of the study. If the subject and/or legal representative decide to withdraw or be withdrawn from study participation, they may request in writing that the study data and samples be destroyed. Subject names or other directly identifiable information will not appear on any reports, publications, or other disclosures of clinical study outcomes.

Clinical data recorded on the electronic database will include intraoperative obstetrician case report forms completed by the obstetrician at the end of surgery, and hospital postpartum morphine equivalent dosing.

#### 10 Adverse Events and Serious Adverse Events

The proposed clinical trial will use the FDA definition of an adverse event (AE). Adverse event means any untoward medical occurrence associated with the use of a drug in humans, whether considered drug related.

The proposed clinical trial will use the FDA definition of SAE. A serious adverse event is any untoward clinical event that is thought by either the investigator or the sponsor to be *unexpected and at least possibly related* to the study and results in any of the following:

- 1. Death
- 2. A life-threatening adverse event
- 3. Inpatient hospitalization or prolongation of an existing hospitalization
- 4. A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- 5. A congenital anomaly or birth defect
- 6. Important medical events that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient, or subject, and may require medical, or surgical intervention to prevent one of the serious outcomes listed above.

Adverse events will be assessed on each participant at stated intervals in Figure 2 section 1.1, both during infusion, and for 12 hours after infusion discontinuation. Duration of monitoring is based on known pharmacokinetics of ketamine.

When an adverse event is discovered, the event will be assessed for severity, relatedness, and expectedness. All adverse events will be documented in the research records and followed until resolved or back to baseline grade.

#### 10.1 Severity

The severity of adverse changes in physical signs or symptoms will be classified as follows:

- *Grade 1 (Mild):* asymptomatic or mild symptoms; clinical or diagnostic observation only; intervention not indicated.
  - e.g., sedation, dizziness, lightheadedness, bad dreams, hallucinations, euphoria, dysphoria, nausea, vomiting
- *Grade 2 (Moderate):* minimal, local, or noninvasive intervention indicated; limiting ageappropriate ADL.
  - o e.g., dysphoria, vomiting
- *Grade 3 (Severe):* medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care/ADL.
  - o e.g., hypertensive urgency or emergency requiring escalated or inpatient treatment
- *Grade 4 (Life-threatening):* consequences; urgent intervention indicated.
  - o e.g., stroke from uncorrected severe hypertension

• *Grade 5 (Death):* event is a direct cause of death.

An independent DSMB will define frequency of monitoring of the tolerability and DLT data.

#### 10.2 Relatedness

Adverse Events and Serious Adverse Events will be subject to the following criteria to determine the relatedness of the experienced event to the research study, protocol, and/or drug.

- Definitely Related There is clear evidence to suggest a causal relationship, and other possible
  contributing factors can be ruled out. The clinical event occurs in a plausible time relationship to
  study intervention administration and cannot be explained by concurrent disease or other drugs or
  chemicals. The response to withdrawal of the drug is clinically plausible. The event must be
  pharmacologically or phenomenologically definitive.
- Probably Related There is evidence to suggest a causal relationship, and the influence of other
  factors is unlikely. The clinical event occurs within a reasonable time after administration of the
  study intervention, is unlikely to be attributed to concurrent disease or other drugs or chemicals
  and follows a clinically reasonable response on withdrawal of the study drug.
- Possibly Related There is some evidence to suggest a causal relationship (e.g., the event occurred within a reasonable time after administration of the study medication). However, other factors may have contributed to the event (e.g., the participant's clinical condition, other concomitant events). Although an AE may rate only as "possibly related" soon after discovery, it can be flagged as requiring more information and later be upgraded to "probably related" or "definitely related", as appropriate.
- Unlikely to be related A clinical event whose temporal relationship to study intervention
  administration makes a causal relationship improbable (e.g., the event did not occur within a
  reasonable time after administration of the study intervention) and in which other drugs or
  chemicals or underlying disease provides plausible explanations (e.g., the participant's clinical
  condition, other concomitant treatments).
- Not Related The AE is completely independent of study intervention administration, and/or evidence exists that the event is related to another etiology. There will be an alternative, definitive etiology documented by the clinician.

#### 10.3 Expectedness

The Principal Investigator will be responsible for determining whether an AE is expected or unexpected. An AE will be considered unexpected if the nature, severity, or frequency of the event is not consistent with the information previously described (sections 8.2 and 9.1). Note that the risks listed in Section 8.1 are considered expected and would <u>not</u> require reporting *unless* the frequency or severity is greater than expected. Events not listed in Section 8.1 but that are listed in the FDA-approved package insert, should

also be considered expected. In such cases, depending on the nature and severity of the event, an amendment may be necessary to add the risk to Section 8.1 and the consent form document.

# 10.4 Reporting Serious Adverse Events

If there is a suggestion that any research procedures have resulted in an injury to subjects, there will be immediate contact with the Principal Investigator who is listed on the first page of the informed consent documents. Any SAE, which is determined by the PI to be unexpected and at least possibly related to study intervention, will be reported to the IRB as soon as possible. The PI is responsible for notifying the FDA within required timeframes. The IDSMB will be notified in writing at the soonest possible timepoint that the event has been identified. The IRB and FDA and will include all known details regarding the nature of the SAE. Outcomes of SAEs not previously reported will be reported to the PI, IRB and FDA via a follow-up report.

Life-threatening or fatal unexpected adverse events associated with the use of the study drug or procedures must be reported to the IRB within 24 hours of discovery of the incident with subsequent follow-up submission of a detailed written report. The IDSMB and IRB will be notified by telephone or facsimile transmission of a human adverse event that is fatal or life-threatening no later than 7 calendar days after receiving the respective human adverse event information, followed by the subsequent submission of a written IND Safety Report. Serious and unexpected adverse events associated with the use of the study drug or procedures will be reported to the IRB with subsequent follow-up submission of a detailed written report in accordance with the respective policies and procedures of the IRB. A summary report of the findings will be prepared and submitted to the regulatory agencies. A written IND Safety Report (i.e., Form FDA 3500A) will be submitted to the FDA as soon as possible and, in no event, later than 15 calendar days following the investigator-sponsor's receipt of the respective adverse event information.

A summary of the SAEs that occurred during the previous year will be included in the FDA annual progress report as well as in the annual IRB continuing review.

# 11 Withdrawal of Subjects and Stopping Rules

This section outlines the criteria that specify when dosing an individual subject, cohort, or trial will be suspended.

#### 11.1 Adverse Events Requiring Discontinuation

For this study, a serious adverse event is any untoward clinical event that is thought by either the investigator or the sponsor to be related to the study and results in any of the following outcomes:

- 1. Death
- 2. A life-threatening adverse event
- 3. Inpatient hospitalization or prolongation of an existing hospitalization

- 4. A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- 5. A congenital anomaly or birth defect
- 6. Important medical events that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient, or subject, and may require medical, or surgical intervention to prevent one of the serious outcomes listed above.

If clinically important and unexpected adverse experiences or clinically important study-related adverse experiences occur, they will be recorded on the adverse event case report form.

Adverse Events Reporting Timeline is documented in 10.4.

# Withdrawal of Subjects due to Adverse Events

Participants will be withdrawn if they experience a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or other important medical events that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient, or subject, and may require medical, or surgical intervention to prevent one of the serious outcomes listed above.

DSMB will review all events pertaining to participant withdrawals. An independent decision will be made regarding trial discontinuation based on risk assessment for current and future trial participants.

Withdrawn participants will be replaced at a proportion of 1:1. Procedures are as follows:

- Study personnel, investigators, and pharmacy will be informed of the need for replacement due to participant withdrawal.
- Subsequent data to be collected from the withdrawn participant will be restricted to the
  minimum amount necessary to continue to monitor safety, i.e., side effect diary including
  questions of sedation, LSD short form, dizziness, lightheadedness, bad dreams, nausea,
  vomiting, pruritus, hallucinations.

# 11.2 Other Criteria Requiring Discontinuation

Withdrawal of Subjects for reasons other than Non-compliance or Adverse Events:

- Protocol non-adherence: incorrect dosing strategy or other non-adherence points at the judgement of the PI
- Incomplete side effect diary data, defined as missing 20% or more responses

Withdrawn participants will be replaced at a proportion of 1:1. Procedures are as follows:

• Study personnel, investigators, DSMB will be informed of the need for replacement due to participant withdrawal.

Subsequent data to be collected from the withdrawn participant will be restricted to the
minimum amount necessary to continue to monitor safety, i.e., side effect diary including
questions of sedation, LSD short form, dizziness, lightheadedness, bad dreams, nausea,
vomiting, pruritus, hallucinations.

## 11.3 Clinical Trial Stopping Rules

This study may be suspended, or prematurely terminated if there is sufficient reasonable cause. DSMB will review all events pertaining to participant withdrawals. An independent decision will be made regarding trial discontinuation based on risk assessment for current and future trial participants.

Written notification, documenting the reason for study suspension or termination, will be provided by the suspending, or terminating party to study participants, investigators, funding agency, the IND sponsor, and regulatory authorities. If the study is prematurely terminated or suspended, the PI will promptly inform study participants, the IRB, and sponsor and will provide the reason(s) for the termination or suspension. Study participants will be contacted, as applicable, and be informed of changes to the study visit schedule.

Circumstances that may warrant termination or suspension include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to participants
- Demonstration of efficacy that would warrant stopping
- Insufficient compliance to protocol requirements
- Data that are not sufficiently complete and/or evaluable
- Determination that the primary endpoint has been met
- Determination of futility

Study may resume once concerns about safety, protocol compliance, and data quality are addressed, and satisfy the sponsor, IRB and/or FDA.

# 12 Statistical Analysis

By virtue of its design, the maximum tolerated dose (MTD) 3+3 design encompasses a minimum number of 6 and maximum number of 12 patients enrolled in this trial. The results identify the drug dose at which ≥33% of patients experience dose limiting toxicity, which we have defined by unacceptable side effects or adverse events. The number of subjects at each dose is dictated by traditional MTD 3+3 design, balancing the risks associated with the study drug and the assessment of adverse event rates. A formal power calculation was not performed.

# 12.1 General Approach

The outcome of this design is the determination of the Maximum Tolerable Dose of ketamine infusion post-cesarean delivery. As such, the final dosing of the MTD design is the primary outcome determined as patient report of tolerated dose and acceptable side effect experiences in greater than 66% of patients.
#### 12.2 Sample Size Determination

The number of subjects (minimum of 6; maximum of 12) at each dose is dictated by traditional MTD 3+3 design, balancing the risks associated with the study drug and the assessment of adverse event rates. A formal power calculation was not performed.

# 12.3 Analysis of Primary Endpoint

Maximum Tolerated (Ketamine) Dose (MTD): The MTD will be defined as the dose at which fewer than 33% of patients experience intolerable effects.

Tolerability (dichotomous Yes/No)

- Tolerability (YES) will be defined as: lack of serious adverse events (serious adverse event defined as: severe unresolved hemodynamic effect: systolic blood pressure <80 or >160, heart rate <40 or >120).<sup>33</sup>
- *Lack of Tolerability* will be defined as presence of any serious adverse event (i.e., severe unresolved hemodynamic effect: systolic blood pressure <80 or >160, heart rate <40 or >120).<sup>33</sup>

For this MTD study, rates of the primary endpoint will be reported as numbers and percentages. Rates of blood pressure and heart rate events will be reported as numbers and percentages.

# 12.4 Analysis of Secondary Endpoints

Side effect acceptability ratings will be reported for each side effect reported as numbers and percentages. Examination of patient pain and depression scores in the 12-weeks post cesarean delivery will be explored. The limited sample size of the MTD design precludes definitive conclusions regarding pain and depression. General linear mixed models will be used to assess trends in pain and depression over the peripartum period according to dose exposure. Paired t-tests may be used to assess changes in pain or depression scores from the preterm to postpartum 12-week assessments.

### 13 Data and Safety Monitoring

Monitoring of safety and data quality in the proposed study will be the responsibility of all personnel on the project, with primary responsibility and supervision by the Investigator. An Independent Data and Safety Monitoring Board (IDSMB) will be convened prior to initiation of the studies and administrated by the University of Pittsburgh CTSI. The study will be reviewed a minimum of quarterly in the first year and twice yearly on an annual basis (or more frequently as deemed necessary) by the IDSMB. The IDSMB will determine the actual frequency of meetings and monitoring, including convening of emergency meetings when necessary.

The Institutional Review Board (IRB) will approve the Statement of Informed Consent for the study and provide institutional oversight of data and safety issues. The study protocol will be approved by the IRB prior to recruiting or obtaining consent from any participants.

Each participant will sign the Informed Consent Form described above prior to participating in the study. To ensure participant safety, once participants are enrolled in the study, study staff will immediately report any adverse and serious adverse events to one of the Investigators. The Investigator will, per standardized procedures, report them to the IDSMB and IRB for review.

# 13.1 Data Safety Monitoring Plan

Monitoring of safety and data quality in the proposed study will be the responsibility of all personnel on the project, with primary responsibility and supervision by the Investigator. There will be an evaluation of the progress of the research study, including assessments of data quality, timelines, participant recruitment, accrual, and retention. The Investigator will also review the outcome and adverse event data to determine whether there is any change to the anticipated benefit-to-risk ratio of study participation and whether the study should continue as originally designed or should it be re-evaluated and changed. A summary report of the data and safety monitoring meetings will be provided to the IRB at the time of the continuing review.

Regarding monitoring of data quality and protected health information, all required personnel proposed for this project will have the required human subjects and confidentiality training, which includes information about maintaining data integrity and security. Confidentiality will be guarded using established procedures such as storing data in locked cabinets within locked offices or locked data rooms, electronic data stored behind UPMC/university firewalls and/or use of REDCap with attendant compliance with data safety standards, coding by study identification numbers rather than any personally identifying information to avoid revealing the identity of subjects, and aggregating data across participants. The key linking names and study identification numbers will be kept separately from the data sets with limited access by study personnel. Only study personnel will have access to the data sets on protected servers. Oversight of all aspects of data management will occur with the Investigator.

#### 13.2 Parameters to be Monitored

The following progress will be monitored throughout the course of the research to ensure the safety of subjects as well as the integrity and confidentiality of their data.

- An evaluation of the progress of the research study, including subject recruitment and retention, and an assessment of the timeliness and quality of the data.
- A review of collected data (including adverse events, unanticipated problems, and subject
  withdrawals) to determine whether there is a change to the anticipated benefit-to-risk
  assessment of study participation and whether the study should continue as originally designed,
  should be changed, or should be terminated (see section 10.1).
- An assessment of external factors or relevant information (e.g., pertinent scientific literature reports or therapeutic development, results of related studies) that may have an impact on the safety and study participants or the ethics of the research study.
- A review of study procedures designed to protect the privacy of the research subjects and the confidentiality of their research data.

The severity of adverse changes in physical signs or symptoms were summarized in section 10.1.

# 13.3 Frequency of Monitoring

The Investigator will review subject safety data as it is generated. The Investigator and the research staff will meet on a weekly interval – and more frequently as necessary – to review data coding and capture, documentation and identification of adverse events, complaints or other issues, and subject confidentiality issues. There will be an evaluation of the progress of the research study, including assessments of data quality, timelines, participant recruitment, accrual, and retention. The PI will also review the outcomes and adverse event data to report to IDSMB who will subsequently decide whether there is any change to the anticipated benefit-to-risk ratio of study participation and whether the study should continue as originally designed or should it be re-evaluated and changed.

An Independent Data and Safety Monitoring Board (IDSMB) will be convened prior to initiation of the studies and administrated by the University of Pittsburgh CTSI. The study will be reviewed a minimum of quarterly in the first year and twice yearly on an annual basis (or more frequently as deemed necessary) by the IDSMB. The IDSMB will determine the actual frequency of monitoring meetings, including convening of emergency meetings when necessary.

### 13.4 Clinical Monitoring

In accordance with 21 CFR 312.50 clinical site monitoring will be conducted to ensure that the rights and well-being of trial participants are protected, that the reported trial data are accurate, complete, and that the conduct of the trial is in compliance with current, approved protocol/amendment(s).

### 13.5 Data and Safety Monitoring Board

An Independent Data and Safety Monitoring Board (IDSMB) will be convened prior to initiation of the studies and administrated by the University of Pittsburgh CTSI. The IDSMB will include individuals in the specialties of Anesthesiology, Psychiatry, Neonatology, and Perinatology as such to create a comprehensive review of the study protocol and participants. The study will be reviewed a minimum of quarterly in the first year and twice yearly on an annual basis (or more frequently as deemed necessary) by the IDSMB. The IDSMB will determine the actual frequency of meetings and monitoring, including convening of emergency meetings when necessary.

## 14 Regulatory, Ethical, and Study Oversight

### 14.1 IRB Approval

The PI will obtain, from the University of Pittsburgh IRB, prospective approval of the clinical protocol and corresponding informed consent form(s); modifications to the clinical protocol and corresponding informed consent forms, and advertisements (i.e., directed at potential research subjects) for study recruitment.

The only circumstance in which a deviation from the current IRB-approved clinical protocol/consent form(s) may be initiated in the absence of prospective IRB approval is to eliminate an apparent immediate hazard to the research subject(s). In such circumstances, the Investigator will promptly notify the University of Pittsburgh IRB of the deviation.

The IRB will review and approve the Informed Consent Document for the study and provide institutional oversight of data and safety issues. The study protocol will be approved prior to recruiting or obtaining consent from any participants. Moreover, the study will be reviewed at a minimum of annual basis (or more frequently as deemed necessary) by the IRB committee. Each participant will sign the approved Informed Consent Form prior to participating in the study.

The University of Pittsburgh IRB operates in compliance with FDA regulations at <u>21 CFR Parts 50</u> and <u>21 CFR 56</u>, and in conformance with applicable ICH Guidelines on GCP.

#### 14.2 Informed Consent Procedures

#### Details of Participant Recruitment:

Subjects approached for enrollment in this study are patients being seen during normal clinical care or by study personnel as part of recruitment procedures as follows. Screening will occur by prenatal clinic, or obstetric operating room schedule, or in the labor and delivery suite. After review, potential patients scheduled for elective cesarean delivery will be approached after clinical staff confirm it is appropriate to do so. For scheduled elective cesarean deliveries, participants will be contacted by phone or in person from obstetric clinic, within 0-21 days prior to the scheduled delivery, to disclose eligibility in the study and to assess their desire to speak to the study team to learn more about the study. The anesthesia team will see all patients presenting for cesarean delivery. During this visit, the anesthesia team typically reviews the patient's medical history, explains the anesthetic plan, and obtains consent for anesthesia. In this study, for eligible participants, investigators will also use this visit to explain the availability of the study to the patient meeting eligibility criteria, when the anesthesiology consult occurs. Should the patient wish to hear more, researchers will discuss risks, benefits, and alternatives to study participation. Questions will be answered, and time will be afforded to patients per the Informed consent Procedures outlined below, minimizing risks of coercion or undue influence.

Recruitment will also occur using Pitt+Me (<a href="https://pittplusme.org/">https://pittplusme.org/</a>) and study fliers within the OBGYN clinics at Magee Womens Hospital. Interested individuals will contact the study team directly. Screening

will take place over the phone, and eligible and interested individuals will be approached prior to their standard cesarean delivery care to go through the informed consent process.

#### Informed Consent Procedures.

The consent process will take place virtually or in person in prenatal clinics or in the preoperative holding area on day of surgery, in accordance with our prior study procedures. The informed consent process will begin when the patient has indicated interest in participating in the study. For women with scheduled cesarean delivery, a phone call with the investigator 0-21 days ahead of time will disclose eligibility and to assess their desire to speak to the study team to learn more about the study. Face-to-face (video and audio) virtual informed consent will be permitted if acceptable to both patient and investigator team, and will follow existing procedures, security and protection protocols that are currently used in our other research protocols.

Patients will be offered additional time to consider the study and their desire to participate - the amount of time for them to consider will be determined by the patient herself and individualized to her level of comfort. They will be informed that they do not need to make any decisions in that encounter and will be encouraged to take time to consider and discuss the study with their support persons without the presence of study personnel. Blank informed consent documents and study brochures will be made available to the subjects and their support people, to support their deliberations.

Individuals will be provided with full explanation of study-related goals and procedures. Questions will be answered for the patient as well as their support people. Patients will be given as much time as they desire to read the consent form and materials and ask questions. If desired, patients can take materials home for review and will be consented to participate via videoconferencing software and electronic consent via REDCap.

Informed consent procedures will be followed and written informed consent will be obtained. No elements of informed consent will be waived.

#### 14.3 Protocol Deviations

Clinical research investigators and staff will be familiarized with the study protocol, GCPs, and applicable federal regulations to ensure that the study protocol procedures are followed. When a deviation is perceived to have occurred, the procedure completed will be verified against the study protocol, applicable regulations and relevant GCP principles. Deviations in the study protocol will be identified verbally and in writing to the PI and/or study coordinator as they occur. In addition to deviations noticed during completion of study protocol procedures, deviations may be identified through routine monitoring visits or audits of the clinical research records, as the research team will meet weekly to review the study recruitment, procedures, and retention. All deviations will be verified and presented to the PI for timely assessment and IRB reporting, if warranted. Any deviation, regardless of severity, will be recorded in the Non-compliance/deviation log by the PI or research staff member as they occur. Protocol deviations that do not meet the definition of IRB reporting requirements will be subject to yearly review and evaluation during the continuing review period.

Deviations determined to be reportable to the IRB include Unanticipated Problems involving risk to participants, Serious Non-compliance with study protocol, and/or Continuing Non-compliance of study protocol. The PI will submit all Unanticipated Problems Involving Risks to Human Subjects or Others and incidents of Reportable Non-compliance within 10 working days of the Investigator becoming aware of the Reportable New Information. *Unanticipated Problems involving risk to participants* include adverse medical occurrences that are:

- Unexpected in terms of nature, severity, or frequency; AND
- Related, or possibly related, to a subject's participation in the research; AND
- Places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

Any protocol deviation that results in an Adverse Events which are unexpected, fatal, or life-threatening, and related or possibly Related to the Research Intervention will be immediately reported to the PI, Clinical Research Coordinator, and reported to the IRB within 24 hours of learning of the event. (All other internal Adverse Events that meet the definition of an Unanticipated Problem Involving Risk to Human Subjects or Others will be reported to the IRB within 10 working days of the investigator learning of the event. If an unexpected adverse event occurs, the investigators will reassess the risk to benefit ratio of the study and will submit any modifications necessary to the IRB. At the time of IRB renewal, the PI will submit information about the frequency of monitoring, any relevant information that may influence the safety or ethical conduct of the study, and any conclusions or changes to the study necessary for continuation, modification, or termination of the study.

Reportable incidence of Non-compliance includes any protocol deviation that:

- Significantly adversely affects the safety, rights, or welfare of the research participants; OR
- Significantly compromises the quality or integrity of the research data (i.e., negatively impacts the ability to draw conclusions from the study data); OR
- Represents Continuing Non-compliance (i.e., has been previously reported or represents a pattern of ongoing non-compliance).

Incidents of Non-compliance that do not meet the IRB reporting requirements will be documented in a Non-compliance/deviation log and managed as part of the Data and Safety Monitoring Plan. The Non-compliance/deviation log will be kept throughout the study and the documentation will be made available upon request.

#### 15 References

- 1. Centers for Disease C, Prevention. Prevalence of self-reported postpartum depressive symptoms-17 states, 2004-2005. *MMWR Morb Mortal Wkly Rep.* 2008;57(14):361-366. PMID: 18401239
- 2. Logsdon MC, Wisner KL, Pinto-Foltz MD. The impact of postpartum depression on mothering. *J Obstet Gynecol Neonatal Nurs*. 2006;35(5):652-658. PMID: 16958723
- 3. Wisner KL, Sit DK, McShea MC, et al. Onset timing, thoughts of self-harm, and diagnoses in postpartum women with screen-positive depression findings. *JAMA Psychiatry*. 2013;70(5):490-498. PMID: 23487258
- 4. Lim G, Facco FL, Nathan N, Waters JH, Wong CA, Eltzschig HK. A Review of the Impact of Obstetric Anesthesia on Maternal and Neonatal Outcomes. *Anesthesiology*. 2018;129(1):192-215. PMID: 29561267
- Lim G, Farrell LM, Facco FL, Gold MS, Wasan AD. Labor Analgesia as a Predictor for Reduced Postpartum Depression Scores: A Retrospective Observational Study. *Anesth Analg*. 2018;126(5):1598-1605. PMID: 29239949
- 6. Lim G, Lasorda K, Farrell L, McCarthy A, Facco FL, Wasan A. Obstetric pain correlates with postpartum depression: a pilot prospective observational study. *BMC Pregnancy Childbirth*. 2020;20(1):240. PMID: 32321455
- 7. Bateman BT, Franklin JM, Bykov K, et al. Persistent opioid use following cesarean delivery: patterns and predictors among opioid-naive women. *American Journal of Obstetrics and Gynecology*. 2016;215(3):353 e351-353 e318. PMID: 26996986
- 8. Peahl AF, Dalton VK, Montgomery JR, Lai YL, Hu HM, Waljee JF. Rates of New Persistent Opioid Use After Vaginal or Cesarean Birth Among US Women. *JAMA Netw Open*. 2019;2(7):e197863. PMID: 31348508
- 9. Komatsu R, Carvalho B, Flood PD. Recovery after Nulliparous Birth: A Detailed Analysis of Pain Analgesia and Recovery of Function. *Anesthesiology*. 2017;127(4):684-694. PMID: 28926443
- 10. Jouguelet-Lacoste J, La Colla L, Schilling D, Chelly JE. The use of intravenous infusion or single dose of low-dose ketamine for postoperative analgesia: a review of the current literature. *Pain Med.* 2015;16(2):383-403. PMID: 25530168
- 11. McIntyre RS, Rosenblat JD, Nemeroff CB, et al. Synthesizing the Evidence for Ketamine and Esketamine in Treatment-Resistant Depression: An International Expert Opinion on the Available Evidence and Implementation. *The American Journal of Psychiatry*. 2021;178(5):383-399. PMID: 33726522
- 12. Lim G, LaSorda KR, Farrell LM, McCarthy AM, Facco FL, Wasan AD. Obstetric pain correlates with postpartum depression symptoms: a pilot prospective observational study. *BMC Pregnancy Childbirth* 2020;20(1):240. PMID: 32321455
- 13. Lim G, LaSorda KR, Rosario B, Krans E, Caritis S. Associations between Postpartum Pain Type with Pain Intensity and Opioid Use in Patients with and without Opioid Use Disorder. *British Journal of Anaesthesia*. 2022;Accepted. PMID: 36371258
- 14. Rajabaliev E, LaSorda K, Ibarra A, Kenkre T, Levine MD, Lim G. Association between labor and delivery pain and postpartum pain with symptoms and clinical diagnosis of postpartum depression in patients with overweight and obesity. *Arch Gynecol Obstet*. 2022. PMID: 35665850

- 15. Abuhelwa AY, Somogyi AA, Loo CK, Glue P, Barratt DT, Foster DJR. Population Pharmacokinetics and Pharmacodynamics of the Therapeutic and Adverse Effects of Ketamine in Patients With Treatment- Refractory Depression. *Clin Pharmacol Ther*. 2022;112(3):720-729. PMID: 35560226
- 16. Li Q, Wang S, Mei X. A single intravenous administration of a sub-anesthetic ketamine dose during the perioperative period of cesarean section for preventing postpartum depression: A meta-analysis. *Psychiatry Research*. 2022;310:114396. PMID: 35278826
- 17. Ma JH, Wang SY, Yu HY, et al. Prophylactic use of ketamine reduces postpartum depression in Chinese women undergoing cesarean section(☆). *Psychiatry Research*. 2019; 279: 252-258. PMID: 31147085
- 18. Yao J, Song T, Zhang Y, Guo N, Zhao P. Intraoperative ketamine for reduction in postpartum depressive symptoms after cesarean delivery: A double-blind, randomized clinical trial. *Brain and Behavior*. 2020;10(9):e01715. PMID: 32812388
- 19. Loo CK, Galvez V, O'Keefe E, et al. Placebo-controlled pilot trial testing dose titration and intravenous, intramuscular and subcutaneous routes for ketamine in depression. *Acta psychiatrica Scandinavica*. 2016;134(1):48-56. PMID: 27028832
- Sultan P, Ando K, Elkhateb R, et al. Assessment of Patient-Reported Outcome Measures for Maternal Postpartum Depression Using the Consensus-Based Standards for the Selection of Health Measurement Instruments Guideline: A Systematic Review. *JAMA Netw Open*. 2022;5(6):e2214885. PMID: 35749118
- 21. Center for Disease Control and Prevention. Prevalence of self-reported postpartum depressive symptoms-17 states, 2004–2005. 2008. PMID: 18401329
- 22. M OH, A S. Rates and risk of postpartum depression-A meta-analysis. *Int Rev Psychiatry*. 1996;8:37-54. PMID: 24211712
- 23. R. S, C. W, V. R, E. S. Moderate to severe depressive symptoms among adolescent mothers followed four years postpartum. . 2006;38:712-718. PMID: 16730600
- 24. K G, C W, A R-G, P D. Correlates of self-reports of being very depressed in the months after delivery: results from the Pregnancy Risk Assessment Monitoring System. *Matern Child Health J.* 2002;6:247-253. PMID: 12512766
- 25. T P, M H, A S, C Z. Postpartum depression. *Am J Obstet Gynecol* 2009;200:357-364. PMID: 19318144
- 26. KP H, CY M. Postpartum Major Depression. *Am Fam Physician*. 2010;81(926-933). PMID: 20949886
- 27. K W, M SDM, D R, et al. Onset timing, thoughts of self-harm, and diagnoses in postpartum women with screen-positive depression findings. *JAMA Psychiatry*. 2013;70(490-8). PMID: 23487258
- 28. V L, JL P, L. C. Prevalence of suicidality during pregnancy and the postpartum. . *Arch Womens Ment Health*. 2005;8:77-87. PMID: 15883651
- 29. Davalos D YC, Tregellas H. Untreated prenatal maternal depression and the potential risks to offspring: a review. . *Arch Womens Ment Health*. 2012;115:1-14. PMID: 22215285
- 30. Murray L AA, Fearon P, Halligan S, Goodyer I, Cooper P. Maternal postnatal depression and the development of depression in offspring up to 16 years of age. . *J Am Acad Child Adolesc Psychiatry*. 2011;50:460-470. PMID: 21515195

- 31. Pearson R EJ, Kounali D, Lewis G, Heron J, Ramchandani P. Maternal depression during pregnancy and the postnatal period: risks and possible mechanisms for offspring depression at age 18 years. *JAMA Psychiatry*. 2013;70:1312-1319. PMID: 24108418
- 32. Micallef J, Tardieu S, Gentile S, et al. Effects of a subanaesthetic dose of ketamine on emotional and behavioral state in healthy subjects. *Neurophysiol Clin.* 2003;33(3):138-147. PMID: 12909392
- 33. Wan LB, Levitch CF, Perez AM, et al. Ketamine safety and tolerability in clinical trials for treatment- resistant depression. *J Clin Psychiatry*. 2015;76(3):247-252. PMID: 25271445
- 34. Hebert MF, Easterling TR, Kirby B, et al. Effects of pregnancy on CYP3A and P-glycoprotein activities as measured by disposition of midazolam and digoxin: a University of Washington specialized center of research study. *Clin Pharmacol Ther*. 2008;84(2):248-253. PMID: 18288078
- 35. Wisner KL, Moses-Kolko EL, Sit DK. Postpartum depression: a disorder in search of a definition. *Arch Womens Ment Health.* 2010;13(1):37-40. PMID: 20127453
- 36. Booth JL, Harris LC, Eisenach JC, Pan PH. A Randomized Controlled Trial Comparing Two Multimodal Analgesic Techniques in Patients Predicted to Have Severe Pain After Cesarean Delivery. *Anesth Analg.* 2016;122(4):1114-1119. PMID: 25806400
- 37. Booth JL, Sharpe EE, Houle TT, et al. Patterns of recovery from pain after cesarean delivery. *Pain*. 2018;159(10):2088-2096. PMID: 29905650
- 38. Eisenach JC, Pan P, Smiley RM, Lavand'homme P, Landau R, Houle TT. Resolution of pain after childbirth. *Anesthesiology*. 2013;118(1):143-151. PMID: 23249931
- 39. Houle TT, Miller S, Lang JE, et al. Day-to-day experience in resolution of pain after surgery. *Pain*. 2017;158(11):2147-2154. PMID: 28708763
- 40. Sharpe EE, Booth JL, Houle TT, et al. Recovery of physical activity after cesarean delivery and its relationship with pain. *Pain.* 2019;160(10):2350-2357. PMID: 31145215
- 41. Carvalho B, Butwick AJ. Postcesarean delivery analgesia. *Best Practice & Research Clinical Anaesthesiology*. 2017;31(1):69-79. PMID: 28625307
- 42. Lavoie A, Toledo P. Multimodal postcesarean delivery analgesia. *Clinics in Perinatology*. 2013;40(3):443-455. PMID: 23972750
- 43. Sutton CD, Carvalho B. Optimal Pain Management After Cesarean Delivery. *Anesthesiology Clinics*. 2017;35(1):107-124. PMID: 28131114
- 44. Verstraete S, Van de Velde M. Post-cesarean section analgesia. *Acta anaesthesiologica Belgica*. 2012;63(4):147-167. PMID: 23610853
- 45. Prabhu M, McQuaid-Hanson E, Hopp S, et al. A Shared Decision-Making Intervention to Guide Opioid Prescribing After Cesarean Delivery. *Obstet Gynecol.* 2017;130(1):42-46. PMID: 28594762
- 46. Badreldin N, Grobman WA, Chang KT, Yee LM. Opioid prescribing patterns among postpartum women. *American Journal of Obstetrics and Gynecology*. 2018;219(1):103.e101-103.e108. PMID: 29630887
- 47. Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. *PloS one*. 2016;11(1):e0147972. PMID: 26824844
- 48. Bateman BT, Cole NM, Maeda A, et al. Patterns of Opioid Prescription and Use After Cesarean Delivery. *Obstet Gynecol*. 2017;130(1):29-35. PMID: 28594763

- 49. Holland E, Bateman BT, Cole N, et al. Evaluation of a Quality Improvement Intervention That Eliminated Routine Use of Opioids After Cesarean Delivery. *Obstet Gynecol.* 2019;133(1):91-97. PMID: 30531571
- 50. Prabhu M, Garry EM, Hernandez-Diaz S, MacDonald SC, Huybrechts KF, Bateman BT. Frequency of Opioid Dispensing After Vaginal Delivery. *Obstet Gynecol.* 2018;132(2):459-465. PMID: 29995732
- 51. Schmidt P, Berger MB, Day L, Swenson CW. Home opioid use following cesarean delivery: How many opioid tablets should obstetricians prescribe? *The Journal of Obstetrics and Gynaecology Research*. 2018;44(4):723-729. PMID: 29359386
- 52. Osmundson SS, Raymond BL, Kook BT, et al. Individualized Compared With Standard Postdischarge Oxycodone Prescribing After Cesarean Birth: A Randomized Controlled Trial. *Obstet Gynecol.* 2018;132(3):624-630. PMID: 30095773
- 53. Osmundson SS, Schornack LA, Grasch JL, Zuckerwise LC, Young JL, Richardson MG. Postdischarge Opioid Use After Cesarean Delivery. *Obstet Gynecol.* 2017;130(1):36-41. PMID: 28594766
- 54. McNicol ED, Midbari A, Eisenberg E. Opioids for neuropathic pain. *The Cochrane Database of Systematic Reviews*. 2013(8):CD006146. PMID: 23986501
- 55. Eisenberg E, McNicol ED, Carr DB. Efficacy and safety of opioid agonists in the treatment of neuropathic pain of nonmalignant origin: systematic review and meta-analysis of randomized controlled trials. *JAMA*. 2005;293(24):3043-3052. PMID: 15972567
- 56. Ballantyne JC, Shin NS. Efficacy of opioids for chronic pain: a review of the evidence. *The Clinical Journal of Pain*. 2008;24(6):469-478. PMID: 18574357
- 57. Chou R, Fanciullo GJ, Fine PG, et al. Clinical guidelines for the use of chronic opioid therapy in chronic noncancer pain. *J Pain*. 2009;10(2):113-130. PMID: 19187889
- 58. Manchikanti L, Kaye AM, Knezevic NN, et al. Responsible, Safe, and Effective Prescription of Opioids for Chronic Non-Cancer Pain: American Society of Interventional Pain Physicians (ASIPP) Guidelines. *Pain Physician*. 2017;20(2s):S3-s92. PMID: 28226332
- 59. Bandura A, O'Leary A, Taylor CB, Gauthier J, Gossard D. Perceived self-efficacy and pain control: opioid and nonopioid mechanisms. *J Pers Soc Psychol*. 1987;53(3):563-571. PMID: 2821217
- 60. Lim G, LaSorda KR, Krans E, Rosario BL, Wong CA, Caritis S. Associations between postpartum pain type, pain intensity and opioid use in patients with and without opioid use disorder: a cross-sectional study. *Br J Anaesth*. 2022;S0007-0912(22):00570-00570. PMID: 36371258
- 61. Wang J, Echevarria GC, Doan L, et al. Effects of a single subanaesthetic dose of ketamine on pain and mood after laparoscopic bariatric surgery: A randomised double-blind placebo controlled study. *Eur J Anaesthesiol*. 2019;36(1):16-24. PMID: 30095550
- 62. Alnefeesi Y, Chen-Li D, Krane E, et al. Real-world effectiveness of ketamine in treatment-resistant depression: A systematic review & meta-analysis. *Journal of Psychiatric Research*. 2022;151:693-709. PMID: 35688035
- 63. Bahji A, Zarate CA, Vazquez GH. Efficacy and safety of racemic ketamine and esketamine for depression: a systematic review and meta-analysis. *Expert Opinion on Drug Safety*. 2022:1-14. PMID: 35231204

- 64. Milak MS, Rashid R, Dong Z, et al. Assessment of Relationship of Ketamine Dose With Magnetic Resonance Spectroscopy of Glx and GABA Responses in Adults With Major Depression: A Randomized Clinical Trial. *JAMA Netw Open.* 2020;3(8):e2013211. PMID: 32785636
- 65. Murrough JW, Iosifescu DV, Chang LC, et al. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. *The American Journal of Psychiatry*. 2013;170(10):1134-1142. PMID: 23982301
- 66. Bauchat JR, Higgins N, Wojciechowski KG, McCarthy RJ, Toledo P, Wong CA. Low-dose ketamine with multimodal postcesarean delivery analgesia: a randomized controlled trial. *International Journal of Obstetric Anesthesia*. 2011;20(1):3-9. PMID: 21224020
- 67. Suppa E, Valente A, Catarci S, Zanfini BA, Draisci G. A study of low-dose S-ketamine infusion as "preventive" pain treatment for cesarean section with spinal anesthesia: benefits and side effects. *Minerva Anestesiol.* 2012;78(7):774-781. PMID: 22374377
- 68. Bilgen S, Koner O, Ture H, Menda F, Ficicioglu C, Aykac B. Effect of three different doses of ketamine prior to general anaesthesia on postoperative pain following Caesarean delivery: a prospective randomized study. *Minerva Anestesiol*. 2012;78(4):442-449. PMID: 22240615
- 69. Heesen M, Bohmer J, Brinck EC, et al. Intravenous ketamine during spinal and general anesthesia for caesarean section: systematic review and meta-analysis. *Acta Anaesthesiol Scand*. 2015;59(4):414-426. PMID: 25789942
- 70. Joel S, Joselyn A, Cherian VT, Nandhakumar A, Raju N, Kaliaperumal I. Low-dose ketamine infusion for labor analgesia: A double-blind, randomized, placebo controlled clinical trial. *Saudi journal of anaesthesia*. 2014;8(1):6-10. PMID: 24665232
- 71. Menkiti ID, Desalu I, Kushimo OT. Low-dose intravenous ketamine improves postoperative analgesia after caesarean delivery with spinal bupivacaine in African parturients. *International Journal of Obstetric Anesthesia*. 2012;21(3):217-221. PMID: 22658477
- 72. Reza FM, Zahra F, Esmaeel F, Hossein A. Preemptive analgesic effect of ketamine in patients undergoing elective cesarean section. *The Clinical Journal of Pain*. 2010;26(3):223-226. PMID: 20173436
- 73. Sen S, Ozmert G, Aydin ON, Baran N, Caliskan E. The persisting analgesic effect of low-dose intravenous ketamine after spinal anaesthesia for caesarean section. *Eur J Anaesthesial*. 2005;22(7):518-523. PMID: 16045141
- 74. Clements JA, Nimmo WS, Grant IS. Bioavailability, pharmacokinetics, and analgesic activity of ketamine in humans. *Journal of Pharmaceutical Sciences*. 1982;71(5):539-542. PMID: 7097501
- 75. Domino EF, Zsigmond EK, Domino LE, Domino KE, Kothary SP, Domino SE. Plasma levels of ketamine and two of its metabolites in surgical patients using a gas chromatographic mass fragmentographic assay. *Anesth Analg.* 1982;61(2):87-92. PMID: 7198883
- 76. Loftus RW, Yeager MP, Clark JA, et al. Intraoperative ketamine reduces perioperative opiate consumption in opiate-dependent patients with chronic back pain undergoing back surgery. *Anesthesiology*. 2010;113(3):639-646. PMID: 20693876
- 77. Vadivelu N, Schermer E, Kodumudi V, Belani K, Urman RD, Kaye AD. Role of ketamine for analgesia in adults and children. *Journal of Anaesthesiology, Clinical Pharmacology*. 2016;32(3):298-306. PMID: 27625475
- 78. Schwenk ES, Viscusi ER, Buvanendran A, et al. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional

- Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. *Reg Anesth Pain Med.* 2018;43(5):456-466. PMID: 29870457
- 79. Deyama S, Sugano Y, Mori S, et al. Activation of the NMDA receptor-neuronal nitric oxide synthase pathway within the ventral bed nucleus of the stria terminalis mediates the negative affective component of pain. *Neuropharmacology*. 2017; 118: 59-68. PMID: 28284823
- 80. Baron R. Peripheral neuropathic pain: from mechanisms to symptoms. *The Clinical Journal of Pain*. 2000;16(2 Suppl):S12-20. PMID: 10870735
- 81. Castel A, Helie P, Beaudry F, Vachon P. Bilateral central pain sensitization in rats following a unilateral thalamic lesion may be treated with high doses of ketamine. *BMC Veterinary Research*. 2013;9:59. PMID: 23537119
- 82. Kaka U, Saifullah B, Abubakar AA, et al. Serum concentration of ketamine and antinociceptive effects of ketamine and ketamine-lidocaine infusions in conscious dogs. *BMC Veterinary Research*. 2016;12(1):198. PMID: 27612660
- 83. Sunder RA, Toshniwal G, Dureja GP. Ketamine as an adjuvant in sympathetic blocks for management of central sensitization following peripheral nerve injury. *Journal of Brachial Plexus and Peripheral Nerve Injury*. 2008;3:22. PMID: 18950516
- 84. Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. *Pain*. 2011;152(3 Suppl):S2-15. PMID: 20961685
- 85. Gaynes BN, Warden D, Trivedi MH, Wisniewski SR, Fava M, Rush AJ. What did STAR\*D teach us? Results from a large-scale, practical, clinical trial for patients with depression. *Psychiatric Services*. 2009;60(11):1439-1445. PMID: 19880458
- 86. Katalinic N, Lai R, Somogyi A, Mitchell PB, Glue P, Loo CK. Ketamine as a new treatment for depression: a review of its efficacy and adverse effects. *Aust N Z J Psychiatry*. 2013;47(8):710-727. PMID: 23661785
- 87. Fava M, Freeman MP, Flynn M, et al. Double-blind, placebo-controlled, dose-ranging trial of intravenous ketamine as adjunctive therapy in treatment-resistant depression (TRD). *Mol Psychiatry*. 2020;25(7):1592-1603. PMID: 30283029
- 88. FDA Prescribing Information Label, SPRAVATO (esketamine) nasal spray, CIII. Initial US Approval: 1970 (ketamine). Reference number: 4399464. 2019.
- 89. Xu Y, Li Y, Huang X, Chen D, She B, Ma D. Single bolus low-dose of ketamine does not prevent postpartum depression: a randomized, double-blind, placebo-controlled, prospective clinical trial. *Arch Gynecol Obstet*. 2017;295(5):1167-1174. PMID: 28357557
- 90. Anderson PO, Sauberan JB. Modeling drug passage into human milk. *Clin Pharmacol Ther*. 2016;100(1):42-52. PMID: 27060684
- 91. Ito S. Drug therapy for breast-feeding women. *The New England Journal of Medicine*. 2000;343(2):118-126. PMID: 10891521
- 92. PN. B. *Use of the monographs on drugs. Drugs and Human Lactation.* Amsterdam: Elsevier; 1996. *ISBN*: 978-0-444-81981-9
- 93. Pai A. Ketamine. Continuing Education in Anaesthesia, Critical Care & Pain, Volume 7, Number 2, 2007, pp 59-63, doi:10.1093/bjaceaccp/mkm008. PMID: 25886322
- 94. Bell RF, Dahl JB, Moore RA, Kalso E. Peri-operative ketamine for acute post-operative pain: a quantitative and qualitative systematic review (Cochrane review). *Acta Anaesthesiol Scand*. 2005;49(10):1405-1428. PMID: 16223384

- 95. Remerand F, Le Tendre C, Baud A, et al. The early and delayed analgesic effects of ketamine after total hip arthroplasty: a prospective, randomized, controlled, double-blind study. *Anesth Analg.* 2009;109(6):1963-1971. PMID: 19923527
- 96. Subramaniam K, Subramaniam B, Steinbrook RA. Ketamine as adjuvant analgesic to opioids: a quantitative and qualitative systematic review. *Anesth Analg.* 2004;99(2):482-495, table of contents. PMID: 15271729
- 97. Corriger A, Voute M, Lambert C, Pereira B, Pickering G, Consortium O. Ketamine for refractory chronic pain: a 1-year follow-up study. *Pain*. 2022;163(4):690-701. PMID: 34252909
- 98. Wang J, Sun Y, Ai P, et al. The effect of intravenous ketamine on depressive symptoms after surgery: A systematic review. *J Clin Anesth.* 2022;77:110631. PMID: 34971992
- 99. Pang L, Cui M, Dai W, Kong J, Chen H, Wu S. Can Intraoperative Low-Dose R,S-Ketamine Prevent Depressive Symptoms After Surgery? The First Meta-Analysis of Clinical Trials. *Front Pharmacol.* 2020;11:586104. PMID: 33192527
- 100. Clements JA, Nimmo WS. Pharmacokinetics and analgesic effect of ketamine in man. *Br J Anaesth*. 1981;53(1):27-30. PMID: 7459184
- 101. Le Tourneau C, Lee JJ, Siu LL. Dose escalation methods in phase I cancer clinical trials. *Journal of the National Cancer Institute*. 2009;101(10):708-720. PMID: 19436029
- 102. Storer BE. Design and analysis of phase I clinical trials. *Biometrics*. 1989;45(3):925-937. PMID: 2790129
- 103. Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. *BMC Health Serv Res.* 2017;17(1):88. PMID: 28126032
- 104. Ely EW, Truman B, Shintani A, et al. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). *JAMA*. 2003;289(22):2983-2991. PMID: 12799407
- 105. C.A. H, J.E. H. Addiction Research Center Inventory (ARCI): measurement of euphoria and other drug effects. New York: Springer-Verlag; 1987 https://doi.org/10.1007/978-1-4612-4812-5\_24
- 106. O'Quigley J, Zohar S. Experimental designs for phase I and phase I/II dose-finding studies. *Br J Cancer*. 2006;94(5):609-613. PMID: 16434987
- 107. Yu N, Tang X, Wang H. Stepwise Confidence Interval Method for MTD Studies with Binomial Populations. Engineering. 2013; 5: 463-466.**DOI:** 10.4236/eng.2013.510B095
- 108. Kamp J, Olofsen E, Henthorn TK, et al. Ketamine Pharmacokinetics. *Anesthesiology*.2020;133(6):1192-1213. PMID: 32997732
- 109. Hodge LS, Tracy TS. Alterations in drug disposition during pregnancy: implications for drug therapy. *Expert Opin Drug Metab Toxicol*. 2007;3(4):557-571. PMID: 17696806
- 110. Isoherranen N, Thummel KE. Drug metabolism and transport during pregnancy: how does drug disposition change during pregnancy and what are the mechanisms that cause such changes? *Drug Metab Dispos.* 2013;41(2):256-262. PMID: 23328895
- 111. Bustos ML, Zhao Y, Chen H, Caritis SN, Venkataramanan R. Polymorphisms in CYP1A1 and CYP3A5 Genes Contribute to the Variability in Granisetron Clearance and Exposure in Pregnant Women with Nausea and Vomiting. *Pharmacotherapy*. 2016;36(12):1238-1244. PMID: 27809336

- 112. Caritis SN, Bastian JR, Zhang H, et al. An evidence-based recommendation to increase the dosing frequency of buprenorphine during pregnancy. *American Journal of Obstetrics and Gynecology*. 2017;217(4):459.e451-459.e456. PMID: 28669739
- 113. Caritis SN, Hankins G, Hebert M, et al. Impact of Pregnancy History and 17-Hydroxyprogesterone Caproate on Cervical Cytokines and Matrix Metalloproteinases. *American Journal of Perinatology*. 2018;35(5):470-480. PMID: 29141262
- 114. Caritis SN, Hauspurg A, Venkataramanan R, Lemon L. Defining the clinical response to 17-alpha hydroxyprogesterone caproate. *American Journal of Obstetrics and Gynecology*. 2018;219(6):623-625. PMID: 30171841
- 115. Hauspurg A, Lemon LS, Serra AE, Sharma S, Venkataramanan R, Caritis SN. Impact of Obesity on the Rate of Recurrent Spontaneous Preterm Birth in Women Treated with 17-alpha Hydroxyprogesterone Caproate. *American Journal of Perinatology*. 2018;35(9):809-814. PMID: 29294501
- 116. Lemon LS, Naimi A, Caritis SN, Platt RW, Venkataramanan R, Bodnar LM. The Role of Preterm Birth in the Association Between Opioid Maintenance Therapy and Neonatal Abstinence Syndrome. *Paediatric and Perinatal Epidemiology*. 2018;32(2):213-222. PMID: 29372750
- 117. Ryu RJ, Easterling TR, Caritis SN, et al. Prednisone Pharmacokinetics During Pregnancy and Lactation. *Journal of Clinical Pharmacology*. 2018;58(9):1223-1232. PMID: 29733485
- 118. Shah M, Xu M, Shah P, et al. Effect of CYP2C9 Polymorphisms on the Pharmacokinetics of Indomethacin During Pregnancy. *European Journal of Drug Metabolism and Pharmacokinetics*. 2018. PMID: 30159654
- 119. Bastian JR, Chen H, Zhang H, et al. Dose-adjusted plasma concentrations of sublingual buprenorphine are lower during than after pregnancy. *American Journal of Obstetrics and Gynecology*. 2017;216(1):64.e61-64.e67. PMID: 27687214
- 120. Caritis S, Zhao Y, Chen HJ, Venkataramanan R. Pharmacodynamics of transdermal granisetron in women with nausea and vomiting of pregnancy. *American Journal of Obstetrics and Gynecology*. 2016;215(1):93.e91-94. PMID: 26812081
- 121. Costantine MM, Cleary K, Hebert MF, et al. Safety and pharmacokinetics of pravastatin used for the prevention of preeclampsia in high-risk pregnant women: a pilot randomized controlled trial. *American Journal of Obstetrics and Gynecology*. 2016;214(6):720.e721-720.e717. PMID: 26723196
- 122. Kalluri HV, Zhang H, Caritis SN, Venkataramanan R. A physiologically based pharmacokinetic modelling approach to predict buprenorphine pharmacokinetics following intravenous and sublingual administration. *British Journal of Clinical Pharmacology*. 2017;83(11):2458-2473. PMID: 28688108
- 123. Lemon LS, Zhang H, Hebert MF, et al. Ondansetron Exposure Changes in a Pregnant Woman. *Pharmacotherapy*. 2016;36(9):e139-141. PMID: 27374186
- 124. Sharma S, Caritis S, Hankins G, et al. Population pharmacokinetics of 17alpha-hydroxyprogesterone caproate in singleton gestation. *British Journal of Clinical Pharmacology*. 2016;82(4):1084-1093. PMID: 27133963
- 125. Elliott J, Plaat F. Burns associated with epidural analgesia and their prevention. *Int J Obstet Anesth.* 2017;32:89-90. PMID: 28684139

- 126. Jin J, Peng L, Chen Q, et al. Prevalence and risk factors for chronic pain following cesarean section: a prospective study. *BMC Anesthesiology*. 2016;16(1):99. PMID: 27756207
- 127. Kainu JP, Halmesmaki E, Korttila KT, Sarvela PJ. Persistent Pain After Cesarean Delivery and Vaginal Delivery: A Prospective Cohort Study. *Anesth Analg.* 2016;123(6):1535-1545. PMID: 19733050
- 128. Landau R, Bollag L, Ortner C. Chronic pain after childbirth. *International Journal of Obstetric Anesthesia*. 2013;22(2):133-145. PMID: 23477888
- 129. Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. *Pain.* 2008;140(1):87-94. PMID: 18818022
- 130. Makeen M, Farrell L, LaSorda K, et al. Associations between postpartum pain, mood, and maternal- infant attachment and parenting outcomes. *Sci Rep.* 2022;12(1):17814. PMID: 36280697
- 131. Demirci JR, Suffoletto B, Doman J, et al. The Development and Evaluation of a Text Message Program to Prevent Perceived Insufficient Milk Among First-Time Mothers: Retrospective Analysis of a Randomized Controlled Trial. *JMIR mHealth and uHealth*. 2020;8(4):e17328. PMID: 32347815
- 132. Kmiec J, Suffoletto B. Implementations of a text-message intervention to increase linkage from the emergency department to outpatient treatment for substance use disorders. *Journal of Substance Abuse Treatment*. 2019;100:39-44. PMID: 30898326
- 133. Pacella ML, Girard JM, Wright AGC, Suffoletto B, Callaway CW. The Association between Daily Posttraumatic Stress Symptoms and Pain over the First 14-days after Injury: An Experience Sampling Study. *Academic Emergency Medicine: Official Journal of the Society for Academic Emergency Medicine*. 2018. PMID: 29513381
- 134. Suffoletto B, Field M, Chung T. Attentional and approach biases to alcohol cues among young adult drinkers: An ecological momentary assessment study. *Experimental and Clinical Psychopharmacology*. 2020;28(6):649-658. PMID: 31886700
- 135. Suffoletto B, Yanta J, Kurtz R, Cochran G, Douaihy A, Chung T. Acceptability of an Opioid Relapse Prevention Text-message Intervention for Emergency Department Patients. *Journal of Addiction Medicine*. 2017;11(6):475-482. PMID: 28858888
- 136. Lam L, Richardson MG, Zhao Z, Thampy M, Ha L, Osmundson SS. Enhanced discharge counseling to reduce outpatient opioid use after cesarean delivery: a randomized clinical trial. *American Journal of Obstetrics & Gynecology MFM*. 2021;3(1):100286. PMID: 33451618
- 137. Schirle LM, Dietrich MS, Lam L, Stone AL, Bruehl S, Osmundson SS. Accuracy of patient-reported versus real-time electronic postoperative opioid use outcomes. *American Journal of Obstetrics & Gynecology MFM*. 2021;3(4):100347. PMID: 33716134
- 138. Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. *The British Journal of Psychiatry: The Journal of Mental Science*. 1987;150:782-786. PMID: 3651732
- 139. Wisner KL, Parry BL, Piontek CM. Clinical practice. Postpartum depression. *The New England Journal of Medicine*. 2002;347(3):194-199. PMID: 12124409
- 140. Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-

- 36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). *Arthritis Care & Research*. 2011;63 Suppl 11:S240-252. PMID: 22588748
- 141. Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987;30(2):191-197. PMID: 3670870
- 142. Katz J, Melzack R. The McGill Pain Questionnaire. In: Turk D, Melzack R, eds. Handbook of Pain Assessment, Third Edition. New York, NY: Guilford Press; 2011:45.
- 143. Cella D, Riley W, Stone A, et al. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005- 2008. *J Clin Epidemiol*. 2010;63(11):1179-1194. PMID: 20685078
- 144. Revicki DA, Chen WH, Harnam N, et al. Development and psychometric analysis of the PROMIS pain behavior item bank. *Pain*. 2009;146(1-2):158-169. PMID: 19683873
- 145. Askew RL, Cook KF, Keefe FJ, et al. A PROMIS Measure of Neuropathic Pain Quality. *Value Health.* 2016;19(5):623-630. PMID: 27565279
- 146. Crofford LJ. Chronic Pain: Where the Body Meets the Brain. *Transactions of the American Clinical and Climatological Association*. 2015;126:167-183. PMID: 26330672
- 147. Khalili R, Sirati Nir M, Ebadi A, Tavallai A, Habibi M. Validity and reliability of the Cohen 10item Perceived Stress Scale in patients with chronic headache: Persian version. *Asian Journal of Psychiatry*. 2017;26:136-140. PMID: 28483077
- 148. Marki G, Bokor A, Rigo J, Rigo A. Physical pain and emotion regulation as the main predictive factors of health-related quality of life in women living with endometriosis. *Human Reproduction* (Oxford, England). 2017;32(7):1432-1438. PMID: 28482063
- 149. Moon HJ, Seo JG, Park SP. Perceived stress in patients with migraine: a case-control study. *The Journal of Headache And Pain*. 2017;18(1):73. PMID: 28733942
- 150. Sibille KT, Langaee T, Burkley B, et al. Chronic pain, perceived stress, and cellular aging: an exploratory study. *Molecular Pain*. 2012;8:12. PMID: 22325162
- 151. Condon J, Corkindale C. The assessment of parent-to-infant attachment: Development of a self-report questionnaire instrument. Journal of Reproductive and Infant Psychology. 2007;16(1):57-76.
- 152. Scopesi A. Assessing mother-to-infant attachment: the Italian adaptation of a self-report questionnaire. Journal of Reproductive and Infant Psychology. 2004;22(2):99-109.
- 153. Van Bussel JC, Spitz B, Demyttenaere K. Three self-report questionnaires of the early mother-to-infant bond: reliability and validity of the Dutch version of the MPAS, PBQ and MIBS. *Arch Womens Ment Health*. 2010;13(5):373-384. PMID: 20127128
- 154. Song J, Zhang T, Choy A, Penaco A, Joseph V. Impact of obesity on post-dural puncture headache. *Int J Obstet Anesth.* 2017;30:5-9. PMID: 28012862
- 155. Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain-United States, 2016. *JAMA*. 2016;315(15):1624-1645. PMID: 26977696
- 156. Silverstein RG, Centore M, Pollack A, Barrieau G, Gopalan P, Lim G. Postpartum psychological distress after emergency team response during childbirth. *J Psychosom Obstet Gynaecol*. 2018:1-7. PMID: 30204531
- 157. Latremoliere A, Woolf CJ. Central sensitization: a generator of pain hypersensitivity by central neural plasticity. *J Pain.* 2009;10(9):895-926. PMID: 19712899
- 158. Koltzenburg M, Lundberg L, Torebjork H. Dynamic and static components of mechanical hyperalgesia in human hairy skin. . *Pain.* 1992;51:207-219. PMID: 1484717

- 159. Brandsborg B, Dueholm M, Kehlet H, Jensen TS, Nikolajsen L. Mechanosensitivity before and after hysterectomy: a prospective study on the prediction of acute and chronic postoperative pain. *Br J Anaesth*. 2011;107(6):940-947. PMID: 21890662
- 160. Granot M, Lowenstein L, Yarnitsky D, Tamir A, Zimmer EZ. Postcesarean section pain prediction by preoperative experimental pain assessment. *Anesthesiology*. 2003;98(6):1422-1426. PMID: 12766652
- 161. Backonja MM, Attal N, Baron R, et al. Value of quantitative sensory testing in neurological and pain disorders: NeuPSIG consensus. *Pain*. 2013;154(9):1807-1819. PMID: 23742795
- 162. Graven-Nielsen T, Aspegren Kendall S, Henriksson KG, et al. Ketamine reduces muscle pain, temporal summation, and referred pain in fibromyalgia patients. *Pain.* 2000;85(3):483-491. PMID: 10781923
- 163. Petersen KK, Arendt-Nielsen L, Simonsen O, Wilder-Smith O, Laursen MB. Presurgical assessment of temporal summation of pain predicts the development of chronic postoperative pain 12 months after total knee replacement. *Pain*. 2015;156(1):55-61. PMID: 25599301
- 164. Attal N, Rouaud J, Brasseur L, Chauvin M, Bouhassira D. Systemic lidocaine in pain due to peripheral nerve injury and predictors of response. *Neurology*. 2004;62(2):218-225. PMID: 14745057
- 165. Edwards RR, Dolman AJ, Martel MO, et al. Variability in conditioned pain modulation predicts response to NSAID treatment in patients with knee osteoarthritis. BMC Musculoskeletal Disorders. 2016;17:284. PMID: 27412526
- 166. Edwards RR, Dolman AJ, Michna E, et al. Changes in Pain Sensitivity and Pain Modulation During Oral Opioid Treatment: The Impact of Negative Affect. *Pain Med.* 2016;17(10):1882-1891. PMID: 26933094
- 167. Edwards RR, Dworkin RH, Turk DC, et al. Patient phenotyping in clinical trials of chronic pain treatments: IMMPACT recommendations. *Pain.* 2016;157(9):1851-1871. PMID: 27152687
- 168. Smith SM, Dworkin RH, Turk DC, et al. The Potential Role of Sensory Testing, Skin Biopsy, and Functional Brain Imaging as Biomarkers in Chronic Pain Clinical Trials: IMMPACT Considerations. *J Pain*. 2017;18(7):757-777. PMID: 28254585
- 169. Wasan AD, Alter BJ, Edwards RR, et al. Test-Retest and Inter-Examiner Reliability of a Novel Bedside Quantitative Sensory Testing Battery in Postherpetic Neuralgia Patients. *J Pain.* 2020;21(7-8):858-868. PMID: 31837446
- 170. Forstenpointner J, Ruscheweyh R, Attal N, et al. No pain, still gain (of function): the relation between sensory profiles and the presence or absence of self-reported pain in a large multicenter cohort of patients with neuropathy. *Pain*. 2021;162(3):718-727. PMID: 32868752
- 171. Petersen KK, Vaegter HB, Stubhaug A, et al. The predictive value of quantitative sensory testing: a systematic review on chronic postoperative pain and the analgesic effect of pharmacological therapies in patients with chronic pain. *Pain.* 2021;162(1):31-44. PMID: 32701654
- 172. Grone E, Crispin A, Fleckenstein J, Irnich D, Treede RD, Lang PM. Test order of quantitative sensory testing facilitates mechanical hyperalgesia in healthy volunteers. *J Pain.* 2012;13(1):73-80. PMID: 22208803
- 173. Martinez V, Fletcher D, Bouhassira D, Sessler DI, Chauvin M. The evolution of primary hyperalgesia in orthopedic surgery: quantitative sensory testing and clinical evaluation before and after total knee arthroplasty. *Anesth Analg.* 2007;105(3):815-821. PMID: 17717244

- 174. Rolke R, Baron R, Maier C, et al. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. *Pain.* 2006;123(3):231-243. PMID: 16697110
- 175. Walk D, Sehgal N, Moeller-Bertram T, et al. Quantitative sensory testing and mapping: a review of nonautomated quantitative methods for examination of the patient with neuropathic pain. *Clin J Pain*. 2009;25(7):632-640. PMID: 19692806
- 176. LaSorda KR, Farrell LM, McClain L, Lim G. Quantitative Sensory Testing to Predict Labor Pain and Postpartum Depression. Poster Presentation. International Anesthesiology Research Society and Association of University Anesthetists. Annual Meeting, May 16-21, 2019, Montreal, Quebec Canada (NCT02692404).
- 177. Lasorda KR, Torre B, Alter B, Krans E, Lim G. Quantitative Psychophysical Correlates of Pain in Pregnant Women with Opioid Use Disorder. ANESTHESIOLOGY Annual Meeting. October 8-13 2021, San Diego, California (NCT04888962).
- 178. McClain L, Farrell L, LaSorda K, Pan LA, Peters D, Lim G. Genetic associations of perinatal pain and depression. *Molecular Pain*. 2019;15:1744806919882139. PMID: 31552780
- 179. Eberhard-Gran M, Eskild A, Tambs K, Opjordsmoen S, Samuelsen SO. Review of validation studies of the Edinburgh Postnatal Depression Scale. *Acta psychiatrica Scandinavica*. 2001;104(4):243-249. PMID: 11722298
- 180. Gibson J, McKenzie-McHarg K, Shakespeare J, Price J, Gray R. A systematic review of studies validating the Edinburgh Postnatal Depression Scale in antepartum and postpartum women. *Acta psychiatrica Scandinavica*. 2009;119(5):350-364. PMID: 19298573
- 181. Cox J, Holden J. Perinatal mental health: A guide to the Edinburgh Postnatal Depression Scale (EPDS). Royal College of Psychiatrists. 2003.
- 182. Sanjuan J, Martin-Santos R, Garcia-Esteve L, et al. Mood changes after delivery: role of the serotonin transporter gene. *The British Journal of Psychiatry: The Journal of Mental Science*. 2008;193(5):383-388. PMID: 18978318
- 183. Ververs FF, Voorbij HA, Zwarts P, et al. Effect of cytochrome P450 2D6 genotype on maternal paroxetine plasma concentrations during pregnancy. *Clinical Pharmacokinetics*. 2009;48(10):677-683. PMID: 19743889
- 184. Spinelli MG, Endicott J. Controlled clinical trial of interpersonal psychotherapy versus parenting education program for depressed pregnant women. *The American Journal of Psychiatry*. 2003;160(3):555-562. PMID: 12611838
- 185. Evans J, Heron J, Francomb H, Oke S, Golding J. Cohort study of depressed mood during pregnancy and after childbirth. *BMJ*. 2001;323(7307):257-260. PMID: 11485953
- 186. Mesches G, Ciolino J, Sticka C, et al. Trajectories of Depressive and Anxiety Symptoms Across Pregnancy and Postpartum in Selective Serotonin Reuptake Inhibitor-Treated Women. *Psychiatry Research and Clinical Practice*. 2022;10.1176/appi.prcp.20210034. PMID: 36254188
- 187. Munk-Olsen T, Laursen TM, Pedersen CB, Mors O, Mortensen PB. New parents and mental disorders: a population-based register study. *JAMA*. 2006;296(21):2582-2589. PMID: 17148723
- 188. Wisner KL, Sit DKY, McShea M, et al. Telephone-Based Depression Care Management for Postpartum Women: A Randomized Controlled Trial. *J Clin Psychiatry*. 2017;78(9):1369-1375. PMID: 28796940

- 189. Nylund K, Asparouhov T, Muthen BO. Deciding On The Number of Classes in Latent Class Analysis and Growth Mixture Modeling: A Monte Carlo Sinulation Study. Structural Equation Modeling. 2007;14(4):535-569.
- 190. Curran PJ, Obeidat K, Losardo D. Twelve Frequently Asked Questions About Growth Curve Modeling. *J Cogn Dev.* 2010;11(2):121-136. PMID: 21743795
- 191. MacCallum RC, Kim C, Malarkey WB, Kiecolt-Glaser JK. Studying Multivariate Change Using Multilevel Models and Latent Curve Models. *Multivariate Behav Res.* 1997;32(3):215-253. PMID: 26761610
- 192. Vittinghoff E, Glidden D, Shiboski S, McCulloch C. Regression Methods in Biostatistics: Linear, Logistic, Survival, and Repeated Measures Models. 2nd ed. New York Dordecht Heidelberg London: Springer; 2012.
- 193. Cappelleri JC, Bushmakin AG, Zlateva G, Sadosky A. Pain responder analysis: use of area under the curve to enhance interpretation of clinical trial results. *Pain Pract.* 2009;9(5):348-353. PMID: 19549060
- 194. Barden J, Edwards J, Moore RA, McQuay HJ. Single dose oral diclofenac for postoperative pain. *The Cochrane Database of Systematic Reviews.* 2004(2):Cd004768. PMID: 15106260
- 195. Dionne RA, Bartoshuk L, Mogil J, Witter J. Individual responder analyses for pain: does one pain scale fit all? *Trends in Pharmacological Sciences*. 2005;26(3):125-130. PMID: 15749157
- 196. Lydick E, Epstein RS, Himmelberger D, White CJ. Area under the curve: a metric for patient subjective responses in episodic diseases. *Quality of Life research: An International Journal of Quality of Life Aspects of Treatment, Care and Rehabilitation.* 1995;4(1):41-45. PMID: 7711690
- 197. Raskin P, Klaff L, McGill J, et al. Efficacy and safety of combination therapy: repaglinide plus metformin versus nateglinide plus metformin. *Diabetes Care*. 2003;26(7):2063-2068. PMID: 12832314
- 198. Toms L, McQuay HJ, Derry S, Moore RA. Single dose oral paracetamol (acetaminophen) for postoperative pain in adults. *The Cochrane Database of Systematic Reviews*. 2008(4):Cd004602. PMID: 18843665

# Appendix 1 – Surveys Measures

| Item | Description, Rationale and Evidence |
|---|---|
| Demographic information | Age, gravidity, parity, estimated gestational age at delivery, weight (kg), height (cm), BMI (kg/m²) |
| | Estimated blood volume on day of surgery (calculated by investigator team): |
| | EBV = 65ml x weight (kg) non-obese |
| | EBV = $50$ ml x weight (kg) obese BMI $\ge 30$ |
| | Smoking status (yes/no), number of prior cesarean deliveries, race/ethnicity, highest level of education, and |
| | household income will be self-reported by subjects. These items relate to social correlates of health that are not |
| | otherwise obtainable by surveys. If differences in these characteristics are observed between groups, a regression |
| | model will control for these factors (see statistical analysis plan). |
| Edinburgh Postnatal | The EPDS is self-completed, 10-item scale specifically for women in the perinatal period. It has been shown to be |
| Depression Scale<br>(EPDS) | an effective means of identifying patients at risk for depression138,139. |
| PROMIS Inventories | PROMIS inventories assess core aspects of pain. PROMIS-PI: Pain interference with activities measures external |
| | manifestations of pain including social role participation and pain interference (i.e., pain behavior). They are |
| | valid and reliable for the constructs that they assess (143-145). |
| Pain intensity<br>(numeric rating scale) | This question assesses the somatic pain experience. |
| 0 | Question: Over the last 24 hours, how intense has your pain been? Please rate on the scale below. 0-10 numeric rating scale where 0 is "no intensity at all" and 10 is "the most intense pain I can imagine" |
| Pain unpleasantness (numeric rating scale) | This question assesses the emotional pain experience, the emotional valence of pain. |
| (,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | Question: Over the last 24 hours, how unpleasant has your pain been? Please rate on the scale below 0-10 numeric rating scale where 0 is "not unpleasant at all" and 10 is "the most unpleasant pain I can imagine" |
| McGill Pain | The McGill Pain Questionnaire Short Form measures multiple dimensions of pain experience including sensory |
| Questionnaire, Short | and affective aspects140,141. The instrument is psychometrically sound, valid, reliable, and has good |
| Form (SF-MPQ) | discriminative capacity142. These measures are necessary to better understand the role that these factors play in |
| | pain intensity, quality, and duration. |
| Perceived Stress<br>Scale (PSS) | Psychological stress/distress affects pain, post-operative recovery, and depression. It will be measured in these populations using the validated Perceived Stress Scale. |
| Daily opioid use | Estimated weekly, daily average (avg) and maximum (max) pill use counts |
| | "Over the last week, how many opioid pills have you used every day on average?" "Over the last week, what was the highest number of opioid pills you have needed for pain?" |
| Opioid use (milligram<br>morphine equivalent,<br>MME) | We will measure oxycodone, hydromorphone and morphine (mg) totals in hospital. These medications will be converted to a single variable, milligram morphine equivalent (MME), per information from the Center for Disease Control |

Appendix 2 – Schedule of Perinatal, Surgical, and Infusion-Specific Research Activities

| | | | Study Visit# 1; Day 0—Delivery/Cesarean Surgery -24 hours post-surgery | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Screening & Baseline Measures | screening<br>seline<br>ures | Presurgical Intake T-1 hour If not completed at baseline | Cesarean Surgery | Ketamine Infusion<br>15-45 minutes Post | 12-hour Ketamine Infusion 12-hour post-infusion | | | | | | | | fusion | | |
| | | | Cesarear | | 15<br>Minutes | 30<br>Minutes | Hour 1 | Hour 4 | Hour 6 | Hour 8 | 10Hour | Hour 12 | Hour 16 | Hour 20 | Hour 24 |
| Informed consent | Х | | | | | | | | | | | | | | |
| Demographics and Medical<br>History (inc. Opioid use in<br>hospital) | Х | Х | | | | | | | | | | | | | |
| Concomitant medication review | Х | X | | | | | | | | | | | | | |
| Administer study intervention | | | | X | | | | | | | | | | | |
| Maternal Plasma Samples <sup>a</sup> | | | | | | | Χ | | Χ | | Χ | X | | | |
| Adverse event review b | | | | X | | | | | | | | | | | X |
| Surgical operative survey | | | | Х | | | | | | | | | | | |
| Pain Intensity | Х | X | | | | | | | | | | | | | |
| Pain Unpleasantness | X | X | | | | | | | | | | | | | |
| PROMIS-PI | X | X | | | | | | | | | | | | | |
| EPDS | Х | X | | | | | | | | | | | | | |
| PSS | X | X | | | | | | | | | | | | | |
| SF-MPQ | Х | X | | | | | | | | | | | | | |
| RASS <sup>b</sup> | | | | | Х | Χ | Χ | Х | | X | X | Х | Х | Χ | X |
| Patient Vitals <sup>b</sup> | | X | | Х | X | Х | Χ | Х | Х | Χ | Χ | Х | Χ | Χ | X |
| LSD Short <sup>b</sup> | | | | | Х | Х | Х | Х | | Х | Х | Х | Х | Х | Х |
| Side Effect Diary and Patient<br>Acceptability <sup>b</sup> | | | | | Х | Х | Х | Х | | Х | Х | Х | Х | Х | Х |

<sup>&</sup>lt;sup>a</sup> Maternal Plasma Sampling includes analysis of Ketamine, ketamine metabolites (Nor-Ketamine & DKNK), Ketamine R- & S-isomers, cortisol, prolactin, and CYP3A and CYP2B6 enzymes

b Adverse Events will result in collection of RASS, LSD short form, Patient vitals, Patient Acceptability ratings, and Maternal plasma sampling at any point between infusion start (t = 0) to 24-hours post-infusion start. LSD score of >8 will trigger a notification to staff and investigator to prompt bedside evaluation.

Appendix 3 – Schedule of Postpartum Research Activities

| Procedures All procedures within +/-3 days | Study<br>Visit 2 | Study<br>Visit 3 | Study<br>Visit 4 | Study<br>Visit 5 | Study<br>Visit 6 | Study<br>Visit 7 | Study<br>Visit 8 | Study<br>Visit 9 | Study<br>Visit 10 | Study<br>Visit 11 | Study<br>Visit 12 | Study<br>Visit 13 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day 7 | Day 14 | Day 21 | Day 28 | Day 35 | Day 42 | Day 49 | Day 56 | Day 63 | Day 70 | Day 77 | Day 84 |
| Pain Intensity | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Pain Unpleasantness | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | × | × |
| PROMIS-PI | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| EPDS | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| PSS | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| SF-MPQ | Х | X | X | X | Х | X | X | X | Х | Х | Х | Х |
| Daily opioid use | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |

Appendix 4. Participant Payment per Task

| | | PREPARE 1 | Payment | | |
|---|---|---|---|---|---|
| Patient<br>Tasks | Timing | Payment | Patient<br>Tasks | Timing | Payment |
| Baseline Sur | rveys | | Postpartum Surveys | | |
| Prior to c | lelivery | \$60 | | Week 1 | \$25 |
| | | | | Week 2 | \$25 |
| Infusion Pay | yments | | | Week 3 \$25 | |
| Plasma | Samples (12 | ml of blood) | | Week 4 \$2 | |
| | T 1 hour | \$62.50 | | Week 5 | \$25 |
| Infusion | T 6 hour | \$62.50 | | Week 6 | \$25 |
| nfu | T 10 hour | \$62.50 | | Week 7 | |
| I | T 12 hour | \$62.50 | | Week 8 | \$25 |
| | Total | \$250.00 | | Week 9 | \$25 |
| | | | | Week 10 | \$25 |
| Side Effe | ct Diaries | | | Week 11 | \$25 |
| Infusion | T 1 hour | \$50.00 | | Week 12 | \$25 |
| | T 6 hour | \$50.00 | | | |
| | T 10 hour | \$50.00 | | Total | \$300 |
| I | T 12 hour | \$50.00 | | | |
| | T 16 hour | \$50.00 | | | |
| t-<br>ion | T 20 hour | \$50.00 | | | |
| Post-<br>Infusion | T 24 hour | \$50.00 | | | |
| I | T 12 hour | \$50.00 | GRA | AND TOTAL | \$1,050 |
| | Total | \$400.00 | | | |
| Vital Signs | 6 | | | | |
| | T 1 hour | \$5.00 | | | |
| Infusion | T 6 hour | \$5.00 | | | |
| | T 10 hour | \$5.00 | | | |
| $\Gamma$ | T 12 hour | \$5.00 | | | |
| | T 16 hour | \$5.00 | | | |
| Post-<br>Infusion | T 20 hour | \$5.00 | | | |
| | T 24 hour | \$5.00 | | | |
| | T 12 hour | \$5.00 | | | |
| | Total | \$40.00 | | | |